


## **Statistical Analysis Plan**

#### Version 1.0

TITLE: 99mTc-rhAnnexin V-128 Planar and SPECT Imaging of Apoptosis in Asymptomatic or Previously Symptomatic with Transient Ischemic Attack (TIA) Patients with Carotid Atherosclerotic Plaque

PROTOCOL #: AAA-Annexin-04 v.5.0 dated 02 February 2018

NCT #: NCT02667457

PHASE: Proof of Concept and Phase II study

DATE: Final version 1.0 dated 24 May 2019

DESIGN: Single centre, single dose, controlled vs healthy volunteers study

INVESTIGATIONAL PRODUCT: Kit for the Preparation of Tc-99m Recombinant Human Annexin V-128 for Injection


Version: 01 Page: **2 of 167** 

## **APPROVAL/REVISION HISTORY**

## Autorship/Approval

| Author: | | Date |
|--------------|--------------------------------------------------|------|
| Approved by: | | Date |
| | Advanced Accelerator Application S.A. (Sponsor), | |

## **Revision history**

| Rev. | Name | Date | Note |
|------|-------|------------|------|
| 01 | Final | 24/05/2019 | |

#### Sent to

| Rev | . Name | e-mail | Sent on | Note |
|-----|--------|--------|------------|------|
| 01 | | | 24/05/2019 | |


Version: 01 Page: **3 of 167** 

## 1 Index

| 1 | Index | 3 | |
|---|---|---|---|
| 2 | List of abl | breviations | 11 |
| 3 | Protocol t | title and number | 13 |
| 4 | INFORMA | ATION TAKEN FROM THE PROTOCOL | 14 |
| | 4.1 Study | y objectives | 14 |
| | 4.1.1 Pn<br>4.1.1.1 | imary objectivePrimary hypothesis | |
| | 4.1.2 Se<br>4.1.2.1 | econdary objectiveSecondary hypotheses | |
| | 4.2 Study | y design | 15 |
| | 4.2.1 Stu | udy population | 15 |
| | 4.2.1.1 | Inclusion criteria | 15 |
| | 4.2.1.2 | Exclusion criteria | 15 |
| | 4.2.2 Stu | udy exposure | 16 |
| | 4.3 Meth | ods and procedures | 16 |
| | 4.3.2 Pa | ource of study population<br>Inticipants study identificationudy procedure | 16 |
| | 4.3.3.1 | Baseline assessments | |
| | 4.3.3.2 | Laboratory assessments | 17 |
| | 4.3.3.3 | 99mTc-rhAnnexin V-128 Planar and SPECT Imaging of the Carotid Arterie | s and Aorta and |
| | Image A | Analysis | 18 |
| | 4.3.3.4 | <sup>99m</sup> Tc-rhAnnexin V-128 Radiation Risk Assessment | 19 |
| | 4.3.3.5 | Ultrasound Examination | 19 |
| | 4.3.3.6 | Withdrawal/discontinuation | 19 |
| | | hedule of assessmentsanned sample size | |
| 5 | SUBJECT | T POPULATIONS (ANALYSIS SETS) | 23 |
| | 5.1 Effica | acy | 23 |
| | 5.1.1 Fu | ıll analysis set (FAS) | 23 |

| | | Version. 01 | . 4 01 107 |
|---|---|---|---|
| | 5.1.2 | Per Protocol population (PP) | 23 |
| | 5.2 | Safety set | 23 |
| | 5.3 | Primary population | 23 |
| 6 | STA | ATISTICAL METHODS | 24 |
| | 6.1 | Statistical analysis strategy | 24 |
| | 6.1.1 | General statistical considerations | 24 |
| | 6.1.2 | P Efficacy endpoint(s) | 24 |
| | 6.1 | 1.2.1 Primary endpoint of PoC | 24 |
| | 6.1 | 1.2.2 Primary endpoint of Phase II | 25 |
| | 6.1 | 1.2.3 Secondary endpoints | 25 |
| | 6.1.3 | Safety endpoint(s) | 26 |
| | 6.1 | 1.3.1 Adverse events | 26 |
| | 6.1 | 1.3.2 Clinical laboratory values | 27 |
| | 6.1 | 1.3.3 Vital signs and physical examination | 27 |
| | 6.1.4 | Missing data and outliers | 27 |
| | 6.1 | 1.4.1 Missing data | 27 |
| | 6.1 | 1.4.2 Missing or incomplete dates | 27 |
| | 6.1 | 1.4.3 Outliers | 28 |
| | 6.1.5 | , , | |
| | 6.1.6<br>6.1.7 | | |
| | 6.1.8 | 5 1 | |
| | 6.1.9 | Subject compliance | 29 |
| | | 0 Prior and concomitant medications | |
| | | 1 Derived data | |
| | | 2 Visit windows | |
| | | 4 Pooling of centres | |
| | | 5 Interim analysis | |
| | | 6 Role of independent data monitoring committee (DMC) / interim data review committee | |
| | | 7 Covariates and analysis of subgroups | |
| | | 8 Sensitivity analysis | |
| | | 20 Significance testing and estimation | |
| 7 | | MPUTER SYSTEMS, SOFTWARE AND VALIDATION OF PROGRAMS | |
| • | | | |
| | | Hardware | |
| | 7.2 | Software | 33 |
| | 7.3 | Validation programs | 33 |

| | | | Version: 01 Page: <b>5 of</b> | 167 |
|---|---|---|---|---|
| 8 | СНА | NGES I | FROM PROTOCOL | 34 |
| 9 | REF | ERENC | ES | 35 |
| 10 | DAT | A PRES | SENTATION | 36 |
| 10 | .1 L | Listings | index | 36 |
| 10 | .2 l | Listing t | emplates | 37 |
| 10 | .3 - | Tables i | index | 37 |
| 10 | .4 | Table te | emplates | 40 |
| 10 | .5 F | Figures | index | 40 |
| 10 | | | emplates | |
| 10 | | Ū | al appendix | |
| 11 | | | =S | |
| 11 | .1 \$ | Standar | d listings | 42 |
| Listin | g 16.2 | | Subject Disposition – All Subjects | |
| Listin | g 16.2 | 2.1.2: | Subject Disposition – Study Withdrawals | 44 |
| Listin | g 16.2 | 2.1.3: | Inclusion Criteria | 45 |
| Listin | g 16.2 | 2.1.4: | Exclusion Criteria | 46 |
| Listin | g 16.2 | 2.1.5: | Screening Failures | 47 |
| Listin | g 16.2 | 2.2: | Protocol Deviations and Reasons for Exclusion from the Study Populations | 48 |
| Listin | g 16.2 | 2.4.1: | Demographics | 49 |
| Listin | g 16.2 | 2.4.2: | Carotid Ultrasound | 50 |
| Listin | g 16.2 | 2.4.3: | Medical History and Associated Pathologies | 51 |
| Listin | g 16.2 | 2.4.4/1: | Prior and Concomitant Medications | 52 |
| Listin | g 16.2 | 2.4.4/2: | Prior and Concomitant Medications | 53 |
| Listin | g 16.2 | 2.5.1/1: | Study Drug Administration and Extent of Subject Exposure | 54 |
| Listin | g 16.2 | 2.5.1/2: | Study Drug Administration and Extent of Subject Exposure | 55 |
| Listin | g 16.2 | 2.6.1: | Carotid and Aorta Imaging Assessment | 56 |

| | Version: 01 | Page: <b>6 of 167</b> |
|---|---|---|
| Listing 16.2.6.2: | Carotid and Aorta Imaging Assessment – Uptake | 57 |
| Listing 16.2.7.1/1: | All Adverse Events | 58 |
| Listing 16.2.7.1/2: | All Adverse Events | 59 |
| Listing 16.2.7.1/3: | All Adverse Events | 60 |
| Listing 16.2.7.2/1: | Serious Adverse Events | 61 |
| Listing 16.2.7.2/2: | Serious Adverse Events | 62 |
| Listing 16.2.7.2/3: | Serious Adverse Events | 63 |
| Listing 16.2.7.3/1: | Adverse Events Leading to Withdrawal | 64 |
| Listing 16.2.7.3/2: | Adverse Events Leading to Withdrawal | 65 |
| Listing 16.2.7.3/3: | Adverse Events Leading to Withdrawal | 66 |
| Listing 16.2.7.4/1: | Adverse Events with Outcome Death | 67 |
| Listing 16.2.7.4/2: | Adverse Events with Outcome Death | 68 |
| Listing 16.2.7.4/3: | Adverse Events with Outcome Death | 69 |
| Listing 16.2.8.1/1: | Hematology | 70 |
| Listing 16.2.8.2/1: | Blood Chemistry | 71 |
| Listing 16.2.8.3/1: | Urinalysis | 72 |
| Listing 16.2.8.4: | Immunogenicity | 73 |
| Listing 16.2.9.1: | Pregnancy Test | 74 |
| Listing 16.2.9.2: | Physical Examination | 75 |
| Listing 16.2.9.3/1: | Vital Signs | 76 |
| Listing 16.2.9.3/2: | Vital Signs | 77 |
| 11.2 Standar | rd Tables | 78 |
| Table 14.1.1: | Subject Disposition | 79 |
| Table 14.1.2: | Analysis Populations | 80 |
| Table 14.1.3: | Protocol Deviations | 81 |
| Table 14.1.4.1: | Demographics – FAS Population | 82 |


Page: **7 of 167** 

| Table 14.1.5.1/1: | Carotid Ultrasound – FAS Population | 83 |
|---|---|---|
| Table 14.1.5.1/2: | Carotid Ultrasound – FAS Population | 84 |
| Table 14.1.6.1: | Medical History and Associated Pathologies – Safety Population | 85 |
| Table 14.1.7.1: | Prior Medications or Non-Drug Therapies – Safety Population | 86 |
| Table 14.1.7.2: | Prior and Concomitant Medications or Non-Drug Therapies – Safety Population | 87 |
| Table 14.1.8.1/1: | Study Drug Administration – Safety Population | 88 |
| Table 14.1.8.1/2: | Study Drug Administration – Safety Population | 89 |
| Table 14.1.8.1/3: | Study Drug Administration – Safety Population | 90 |
| Table 14.2.1.1:<br>91 | Carotid and Aorta Imaging Assessment – Prevalence of Positive Scans – FAS Population | on |
| Table 14.2.1.2: 92 | Carotid and Aorta Imaging Assessment – Prevalence of Positive Scans – PP Population | on |
| Table 14.2.1.3:<br>Population | Patient Carotid and Aorta Imaging Assessment – Comparison between time points – FA | ٩S |
| Table 14.2.1.4:<br>Population | Left Carotid Uptake Imaging Assessment – Target to Background Ratio (TBR) – FA | ٩S |
| Table 14.2.1.5:<br>Population | Right Carotid Uptake Imaging Assessment – Target to Background Ratio (TBR) – FA | ٩S |
| Table 14.2.1.6:<br>Population | Thoracic Aorta Uptake Imaging Assessment – Target to Background Ratio (TBR) – FA | ٩S |
| Table 14.2.1.7:<br>Population | Abdominal Aorta Uptake Imaging Assessment – Target to Background Ratio (TBR) – FA | ٩S |
| Table 14.2.1.8:<br>Population | Aortic Arch Uptake Imaging Assessment – Target to Background Ratio (TBR) – FA 98 | ٩S |
| Table 14.2.1.9: echolucency/echo | Left Carotid Uptake Imaging Assessment by ultrasound grade of plaque genicity – Target to Background Ratio (TBR) – Patients - FAS Population | |
| | Right Carotid Uptake Imaging Assessment by ultrasound grade of plaque genicity – Target to Background Ratio (TBR) – Patients - FAS Population | |
| Table 14.3.1.1: | Overall Summary of Adverse Events – Safety Population | 01 |
| Table 14.3.1.2:<br>System Organ Cla | Number (%) of Subjects Reporting Treatment Emergent Adverse Events by Prima ass and Preferred Term – Safety Population | |

Version: 01


Version: 01 Page: **8 of 167** 

| Table 14.3.1.3:<br>Safety Population | Number (%) of Subjects Reporting Treatment Emergent Adverse Events by Seventing 103 | rity – |
|---|---|---|
| Table 14.3.1.4:<br>Severity – Safety F | Number (%) of Subjects Reporting Treatment Emergent Adverse Drug Reaction | - |
| Table 14.3.1.5:<br>Primary System O | Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Event<br>rgan Class and Preferred Term – Safety Population | |
| Table 14.3.1.6:<br>Severity – Safety F | Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Event | |
| Table 14.3.1.7:<br>by Severity – Safe | Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Drug Reactly Population | |
| Table 14.3.2.1: | Listing of Adverse Events with Outcome Death – Safety Population | . 108 |
| Table 14.3.2.2: | Listing of Serious Adverse Events – Safety Population | . 109 |
| Table 14.3.4: | Abnormal Laboratory Value Listing (Each Patient) – Safety Population | . 110 |
| Table 14.3.5.1/1: | Hematology – Red blood cells (10 <sup>12</sup> /L) – Safety Population | . 111 |
| Table 14.3.5.1/2: | Hematology – Hematocrit (L/L) – Safety Population | . 112 |
| Table 14.3.5.1/3: | Hematology – Hemoglobin (g/L) – Safety Population | . 113 |
| Table 14.3.5.1/4: | Hematology – White blood cells (109/L) – Safety Population | . 114 |
| Table 14.3.5.1/5: | Hematology – Basophils (109/L) – Safety Population | . 115 |
| Table 14.3.5.1/6: | Hematology – Eosinophils (10 <sup>9</sup> /L) – Safety Population | . 116 |
| Table 14.3.5.1/7: | Hematology – Lymphocytes (10 <sup>9</sup> /L) – Safety Population | . 117 |
| Table 14.3.5.1/8: | Hematology – Monocytes (10 <sup>9</sup> /L) – Safety Population | . 118 |
| Table 14.3.5.1/9: | Hematology – Neutrophils (10 <sup>9</sup> /L) – Safety Population | . 119 |
| Table 14.3.5.1/10: | Hematology – Platelet Count (109/L) – Safety Population | . 120 |
| Table 14.3.5.1/11: | Hematology – PT (Second) – Safety Population | . 121 |
| Table 14.3.5.1/12: | Hematology – PTT (Second) – Safety Population | . 122 |
| Table 14.3.5.1/13: | Hematology – INR – Safety Population | . 123 |
| | Blood Chemistry – ALP (U/L) – Safety Population | |
| | Blood Chemistry – ALT (U/L) – Safety Population | |
| | Blood Chemistry – AST (II/I ) – Safety Population | 126 |


| | | Blood Chemistry – Total Bilirubin (µmol/L) – Safety Population | |
|---|---|---|---|
| Table | 14.3.5.2/5: | Blood Chemistry – Direct Bilirubin (µmol/L) – Safety Population | 28 |
| Table | 14.3.5.2/6: | Blood Chemistry – Gamma-GT (U/L) – Safety Population | 29 |
| Table | 14.3.5.2/7: | Blood Chemistry – Blood Urea Nitrogen (mmol/L) – Safety Population 1 | 30 |
| Table | 14.3.5.2/8: | Blood Chemistry – Albumin (g/L) – Safety Population | 31 |
| Table | 14.3.5.2/9: | Blood Chemistry – Serum Creatinine (µmol/L) – Safety Population | 32 |
| Table | 14.3.5.2/10: | Blood Chemistry – Uric Acid (µmol/L) – Safety Population | 33 |
| Table | 14.3.5.2/11: | Blood Chemistry – Sodium (mmol/L) – Safety Population | 34 |
| Table | 14.3.5.2/12: | Blood Chemistry – Potassium (mmol/L) – Safety Population | 35 |
| Table | 14.3.5.2/13: | Blood Chemistry – Phosphorus (mmol/L) – Safety Population | 36 |
| Table | 14.3.5.2/14: | Blood Chemistry – Chloride (mmol/L) – Safety Population | 37 |
| Table | 14.3.5.2/15: | Blood Chemistry – Corrected Calcium (mmol/L) – Safety Population | 38 |
| Table | 14.3.5.2/16: | Blood Chemistry – Glucose (mmol/L) – Safety Population | 39 |
| Table | 14.3.5.2/17: | Blood Chemistry – Total Protein (g/L) – Safety Population | 40 |
| Table | 14.3.5.2/18: | Blood Chemistry – LDH (U/L) – Safety Population | 41 |
| Table | 14.3.5.2/19: | Blood Chemistry – Total Cholesterol (mmol/L) – Safety Population | 42 |
| Table | 14.3.5.3/1: | Urinalysis – Blood – Safety Population | 43 |
| Table | 14.3.5.3/2: | Urinalysis – pH – Safety Population | 44 |
| Table | 14.3.5.3/3: | Urinalysis – Specific Gravity – Safety Population | 45 |
| Table | 14.3.5.3/4: | Urinalysis – Protein – Safety Population | 46 |
| Table | 14.3.5.3/5: | Urinalysis – Glucose – Safety Population | 47 |
| Table | 14.3.5.3/6: | Urinalysis – Ketones – Safety Population | 48 |
| Table | 14.3.5.3/7: | Urinalysis – RBC (per high power field) – Safety Population 1 | 49 |
| Table | 14.3.5.3/8: | Urinalysis – WBC (per high power field) – Safety Population 1 | 50 |
| Table | 14.3.5.3/9: | Urinalysis – Casts – Safety Population | 51 |
| Table | 14.3.6.1/1: | Vital Signs – Systolic Blood Pressure (mmHg) – Safety Population 1 | 52 |

Version: 01

| | Version: 01 | Page: <b>10 of 167</b> |
|---|---|---|
| Table 14.3.6.1/2: \ | Vital Signs – Diastolic Blood Pressure (mmHg) – Safety Population | 153 |
| Table 14.3.6.1/3: \ | /ital Signs – Heart Rate (beats/min) – Safety Population | 154 |
| 11.3 Standard | l Figures | 155 |
| | Left Carotid Target to Background Ratio (TBR) Imaging Assessment - P<br>6 – FAS Population - 60 mins after IP injection | |
| | Left Carotid Target to Background Ratio (TBR) Imaging Assessment - P<br>6 – FAS Population - 120 mins after IP injection | |
| | Right Carotid Target to Background Ratio (TBR) Imaging Assessment - F<br>6 – FAS Population - 60 mins after IP injection | |
| | Right Carotid Target to Background Ratio (TBR) Imaging Assessment - F<br>6 – FAS Population - 120 mins after IP injection | |
| | Scatterplot between Left and Right Carotid and Thoracic Aorta Target to E<br>FAS Population - 60 mins after IP injection | |
| | Scatterplot between Left and Right Carotid and Thoracic Aorta Target to E<br>FAS Population - 120 mins after IP injection | |
| | Scatterplot between Left and Right Carotid and Abdominal Aorta Targents – FAS Population - 60 mins after IP injection | |
| Figure 14.2.1.8: S<br>Ratio (TBR) – Patie | Scatterplot between Left and Right Carotid and Abdominal Aorta Targents – FAS Population - 120 mins after IP injection | et to Background |
| | Scatterplot between Left and Right Carotid and Aortic Arch Target to B FAS Population - 60 mins after IP injection | |
| | Scatterplot between Left and Right Carotid and Aortic Arch Target to B FAS Population - 120 mins after IP injection | |
| 12 APPENDICES | S TO THE SAP TEMPLATE | 166 |
| 12.1 Derived of | data | 166 |
| 12.2 SAS prog | grams | 167 |


Version: 01 Page: **11 of 167** 

#### 2 List of abbreviations

AAA Advanced Accelerator Applications

AE Adverse Event

ALAT Alanine Aminotransferase

ALP Alkanine Phosphatase

ALT Alanine Transaminase

ASAT Aspartate Aminotransferase

AST Aspartate Transaminase

ATC Anatomical Therapeutic Chemical classification system

BMI Body Mass Index

BP Blood Pressure

BUN Blood Urea Nitrogen

C.I. Confidence Interval

CRF Case Report Form

CRO Clinical Research Organization

CT Computed Tomography

DMC Data Monitoring Committee

eCRF electronic Case Report Form

FAS Full Analysis Set

GGT Gamma-Glutamyl Transpeptidase

Hb Hemoglobin

HR Heart Rate

ICH International Conference on Harmonization

ID Identification

IP Intraperitoneal

IQR Interquartile Range

kVp Peak Kilovoltage

LDH Lactate Dehydrogenase


Version: 01 Page: **12 of 167** 

LLT Lowest Level Term

MBq Mega Becquerel

MCID Minimal Clinically Important Difference

MCV Mean Corpuscular Volume

MHLTC Ministry of Health and Long Term Care

MedDRA Medical Dictionary for Regulatory Activities

OHSN-REB Ottawa Hospital Science Network Research Ethics Board

PoC Proof of Concept

PP Per Protocol

PT Preferred Term

RBC Red Blood Cell

ROC Receiver Operator Characteristic curve

SAE Serious Adverse Event

SAP Statistical Analysis Plan

S.D. Standard Deviation

SPECT Single Photon Emission Computed Tomography

SOC System Organ Class

TEAEs Treatment emergent Adverse events

VOIs Volumes Of Interest

WBC White Blood Cell






Version: 01 Page: **13 of 167** 

## 3 Protocol title and number

<sup>99m</sup>Tc-rhAnnexin V-128 Planar and SPECT Imaging of Apoptosis in Asymptomatic or Previously Symptomatic with Transient Ischemic Attack (TIA) Patients with Carotid Atherosclerotic Plaque (Protocol Number AAA-Annexin-04 v.5.0 dated 02 February 2018).



Version: 01 Page: **14 of 167** 

#### 4 INFORMATION TAKEN FROM THE PROTOCOL

## 4.1 Study objectives

#### 4.1.1 Primary objective

The primary objective of this investigation is to determine the feasibility of imaging apoptotic activity in carotid atherosclerotic plaques of asymptomatic or previous symptomatic with TIA only patients with significant carotid artery disease by using <sup>99m</sup>Tc-rhAnnexin V-128 imaging and to report the prevalence of abnormal <sup>99m</sup>Tc-rhAnnexin V-128 scans.

#### 4.1.1.1 Primary hypothesis

<sup>99m</sup>Tc-rhAnnexin V-128 imaging can be used to detect apoptosis in carotid plaque in asymptomatic or previously symptomatic with TIA only patients with at least 50% carotid stenosis as defined by ultrasound. In this population, the anticipated prevalence of carotid apoptosis will be 0.3 to 0.5.

#### 4.1.2 Secondary objective

The secondary objectives are:

- To establish the uptake of <sup>99m</sup>Tc-rhAnnexin V-128 in a control group of participants with normal carotid ultrasounds.
- To assess the <sup>99m</sup>Tc-rhAnnexin V-128 uptake versus plaque echogenicity and echolucency.
- To measure aortic uptake of <sup>99m</sup>Tc-rhAnnexin V-128 and assess the correlation with its carotid uptake.

#### 4.1.2.1 Secondary hypotheses

- <sup>99m</sup>Tc-rhAnnexin V-128 uptake will be increased in plaque with greater echogenicity.
- 99mTc-rhAnnexin V-128 uptake will be decreased in plaque with greater echolucency.
- 99mTc-rhAnnexin V-128 imaging can be used to detect apoptosis in the aorta in asymptomatic patients with at least one 50% carotid stenosis as defined by ultrasounds.
- Aortic uptake of <sup>99m</sup>Tc-rhAnnexin V-128 will be correlated with carotid uptake of <sup>99m</sup>Tc-rhAnnexin V-128.



Version: 01 Page: **15 of 167** 

#### 4.2 Study design

This is a single-centre, single dose, Proof of Concept (PoC), Phase II study. Participants will receive a single intravenous bolus of 350 MBq ± 10 % of <sup>99m</sup>Tc-rhAnnexin V-128 followed by SPECT/CT imaging of the carotids and aortas. Carotid plaque echogenicity and echolucency will be assessed by carotid ultrasounds carried out within 8 weeks of <sup>99m</sup>Tc-rhAnnexin V-128 SPECT/CT imaging. SPECT/CT <sup>99m</sup>Tc-rhAnnexin V-128 carotid imaging will be obtained in 35 asymptomatic participants with at least one ≥ 50% carotid stenosis and in 10 participants with normal carotid ultrasounds.

#### 4.2.1 Study population

Approval for the study was obtained from the Ottawa Hospital Science Network Research Ethics Board (OHSN-REB) and Health Canada. All participants will provide written informed consent prior to the initiation of any study procedures. Thirty-five participants with carotid stenosis and ten age and sex matched control participants will be enrolled.

#### 4.2.1.1 Inclusion criteria

For all participants:

- 1. Males and females age 18 years or greater;
- 2. Able and willing to comply with the study procedures;
- 3. Negative pregnancy test for women of childbearing potential at screening and on the day of administration of <sup>99m</sup>Tc-rhAnnexin V-128.

For participants with carotid artery disease:

4. Evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 10 years;

For control participants:

4. No significant carotid artery disease on carotid ultrasound.

#### 4.2.1.2 Exclusion criteria

- 1. Previous carotid stenting or endarterectomy, or stroke;
- 2. Diagnosis of vasculitis, dissection, or non-atherosclerotic carotid disease (Ehlers-Danlos, Marfans);
- 3. Pregnancy or lactation;



Version: 01 Page: **16 of 167** 

- 4. History of any disease or relevant physical or psychiatric condition or abnormal physical finding which may interfere with the study objectives at the investigator judgment;
- 5. Know hypersensitivity to the investigational product or any of its components;
- 6. Claustrophobia or inability to lie still in a supine position;
- 7. Participation in another clinical trial within 4 weeks before study inclusion, except for patients who have participated or who are currently participating in a study without any study drug administration:
- 8. Unwillingness to provide consent.

#### 4.2.2 Study exposure

Subjects will be exposed to only one injection of <sup>99m</sup>Tc-rhAnnexin V-128 for SPECT/CT imaging of the carotids and aortas.

### 4.3 Methods and procedures

#### 4.3.1 Source of study population

The carotid artery study population will be adult male and female patients who are referred to the outpatient cardiology clinics and/or the non-invasive Diagnostic Imaging Department at the University of Ottawa Heart Institute. The control population will be healthy volunteers who do not have carotid atherosclerosis as assessed by ultrasounds and whose lab values are within the normal range.

#### 4.3.2 Participants study identification

Each participant will be identified with a participant ID number. A unique participant identification number (Participant ID) will be assigned at the start of the screening period to each participant who signs the informed consent form. This number will identify the participant throughout the study. Participant IDs will include the 2-digit protocol number (04), the 2-letter code (CA) and a 3- digit participant number (ex: 04-CA-001 for first participant in).

#### 4.3.3 Study procedure

Voluntary written informed consent will be obtained prior to the initiation of any study-related procedures. Study conduct procedures will include a screening visit, the imaging studies, a phone visit within 24 hour post <sup>99m</sup>Tc-rhAnnexin V-128 administration visit and a visit at 30 days.



Version: 01 Page: **17 of 167** 

#### 4.3.3.1 Baseline assessments

- Each participant's date of birth (mm/yyyy), gender, ethnicity, weight, height, medical history, and relevant baseline characteristics will be recorded.
- Results from any standard of care testing related to the participant's condition will be collected.
- Women of childbearing potential must have negative pregnancy test at screening and before the investigational product administration.
- Limited physical exam (height, weight, BMI) and vital signs (systolic and diastolic blood pressure, heart rate), will be recorded.

#### 4.3.3.2 Laboratory assessments

Blood samples for hematology, biochemistry and urinalysis will be obtained at baseline for screening,  $30 \pm 3$  days post IP administration and following any adverse events.

In case of clinically significant abnormalities in baseline laboratory values, the participant will be declared as a screening failure.

| Hematology | Coagulation | Blood Chemistry | Urinalysis |
|---|---|---|---|
| WBC with differential RBC Platelets Hb MCV Hematocrit | • PT<br>• PTT<br>• INR | <ul> <li>BUN</li> <li>Uric Acid</li> <li>Albumin</li> <li>Direct bilirubin</li> <li>LDH</li> <li>Calcium</li> <li>Chloride</li> <li>Phosphorus</li> <li>Total cholesterol</li> <li>Total protein</li> <li>Serum creatinine</li> <li>Total bilirubin</li> <li>ALP</li> <li>AST/ASAT</li> <li>ALT/ALAT</li> <li>Gamma-GT</li> <li>Sodium</li> <li>Potassium</li> <li>Glucose</li> <li>β-HCG at screening</li> </ul> | Dipstick test <sup>1</sup> Pregnancy test (before injection of study product, if applicable) |

<sup>&</sup>lt;sup>1</sup> In case one of the assessments of the dipstick test is positive, a microscopic analysis of the urine must be performed.



Version: 01 Page: **18 of 167** 

Laboratory Assessments will be performed by the ■

The Ottawa Hospital according to Ministry of Health and Long Term Care (MHLTC) standards.

To rule out development of anti-annexin V-128 antibodies, venous blood samples will also be drawn for each participant at screening and 30 ± 3 days post <sup>99m</sup>Tc-rhAnnexin V-128 injection. Assays for anti-rhAnnexin V-128 IgG and IgM antibodies will be performed in serum samples by ELISA. For this purpose, 10 mL of blood will be collected for each assay.

## 4.3.3.3 99mTc-rhAnnexin V-128 Planar and SPECT Imaging of the Carotid Arteries and Aorta and Image Analysis

Planar and SPECT imaging of the carotids and aorta will be performed 60 and 120 minutes after injection of tracer.

Administration of the <sup>99m</sup>Tc-rhAnnexin V-128 (350 MBq ± 10%) will be as a single bolus via an intravenous catheter in an antecubital vein followed by a saline flush. Negative pregnancy test for women of childbearing potential will be confirmed on the day of administration.

All images will be acquired with a dual head SPECT/CT gamma camera with low-energy high-resolution collimators. The energy acceptance window for the <sup>99m</sup>Tc photopeak will be 140 keV (± 10%). A low dose CT scan (helical, 120 kVp, 1 mA with 1.9 pitch) will be acquired of the neck, thorax and abdomen for attenuation correction.

Reconstruction will be done using iterative reconstruction incorporating CT-based attenuation correction and dual-energy-window scatter correction. SPECT images of the carotid arteries and thoracic and abdominal aorta will be acquired at 1 and 2 hours post-injection. Acquired images will be stored for off-line analysis using a Hermes Gold workstation (Hermes Medical Solutions). Volumes-of-interest (VOIs) will be placed over the carotids and the thoracic and abdominal aortic sections to determine image counts from the attenuation and scatter corrected images. A <sup>99m</sup>Tc source of known activity will be imaged and used to determine the imaging system calibration factor for converting reconstructed image counts into an activity concentration (MBq/cc or % injected dose/gram).

A normal database of carotid and aortic uptake will be determined from 10 control participants and used to identify abnormal uptake in carotid artery disease participants.

Inter and intra-observer variability will be determined by repeated analysis of the images of 20 participants. Two observers will carry out the assessment of inter-observer variability. Images will be anonymized prior to analysis and observers will be blinded to all clinical data.





#### 4.3.3.4 99mTc-rhAnnexin V-128 Radiation Risk Assessment

Participants will receive radiation from 1) <sup>99m</sup>Tc-rhAnnexin V-128 (350 MBq) for a dose of 2.2 mSv (7.7 ± 0.8 uSv/MBq) and 2) the CT scan for attenuation correction for a dose of 1.8 mSv. Total dose for <sup>99m</sup>Tc-rhAnnexin V-128 and CT components will be 4.0 mSv.

#### 4.3.3.5 Ultrasound Examination

Clinical evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 10 years prior to enrolment is required for inclusion in the trial.

Evidence of 50% or more carotid stenosis has to be confirmed in a more recent US imaging within 8 weeks prior to <sup>99m</sup>Tc-rhAnnexin V-128 administration. If not confirmed, the participant will be declared as a screening failure.

B-mode and color Doppler ultrasound studies will be acquired of both carotid arteries and performed with an ultrasound scanner equipped with a 5- to 7-MHz transducer. Plaque morphology, as echogenicity, defined as reflectance of the emitted ultrasound signal, will be assessed as previously described and graded from 1 to 4 as echolucent, predominantly echolucent, predominantly echogenic, or echogenic. The vessel lumen will be used as the reference structure for defining echolucency, and the bright echo zone produced by the media-adventitia interface in the far wall will be used as the reference structure for defining echogenicity. Interobserver reproducibility of plaque morphology in stenotic arteries has been previously assessed ( $\kappa$ =0.56, 95% C.I. 0.38 to 0.74).

The degree of stenosis will be calculated by the following equation: (1-PSVr/PSVs)×100%, where PSVr denotes peak systolic velocity at the point of reference (here, the distal carotid artery) and PSVs the peak systolic velocity in the stenosis.

#### 4.3.3.6 Withdrawal/discontinuation

The withdrawal of a study participant is mandatory in the following cases:

- Pregnancy
- Protocol violation determined as critical
- Lost to follow-up
- Serious inter-current illness or other safety reasons for what the Investigator considers it is in the best interest of the participant to withdraw from the study
- Screening failure





A "screening failure" is a participant who has signed the informed consent, but who does not meet all selection criteria following the screening evaluations. For participants not considered eligible after the screening period, the reason for not being eligible must be documented. No additional assessments are needed. Participant information collected at the screening visit will be entered in the eCRF and will be used in the study analysis.

The participants may withdraw from the study if they decide to do so, at any time and irrespective of the reason, or this may be the Investigator's decision. The primary reason for a participant's withdrawal from the study should be determined if possible. The date and reason for discontinuation will be documented in the eCRF.

#### 4.3.4 Schedule of assessments

Participants who have signed the informed consent and are eligible to participate in the study will undergo the following assessments:

- A screening visit will be conducted within 8 weeks prior to the <sup>99m</sup>Tc-rhAnnexin V-128 imaging. Eligible and consenting participants will undergo a limited physical examination (height, weight, BMI), vital signs (systolic and diastolic blood pressure, heart rate), blood analysis and urinalysis. The following blood analysis will be conducted: CBC with automated differential, general chemistry panel (SMA-20) including PT/PTT, INR (international normalized ratio for PT values) and assessment of anti-annexin V-128 antibodies.
- Carotid ultrasound will be carried out within 8 weeks prior to the <sup>99m</sup>Tc-rhAnnexin V-128 SPECT/CT imaging. SPECT Imaging visit: dedicated SPECT/CT imaging of the carotids and aorta will be done 60 minutes after injection of tracer, and 120 minutes after injection. Vital signs assessment/participant monitoring will be done throughout the visit.
- Within 24 hours after the administration of <sup>99m</sup>Tc-rhAnnexin V-128, participants will be called for the assessment of possible adverse events.
- 30 ± 3 days post <sup>99m</sup>Tc-rhAnnexin V-128 injection, all participants will return to clinic for a final blood sampling to rule out the development of anti-annexin V-128 antibodies. The following blood analysis will also be conducted: CBC with automated differential, general chemistry panel (SMA-20) including PT/PTT, and INR.
- Once the first 15 patients and 5 normals have been administered with <sup>99m</sup>Tc-rhAnnexin V-128 and have performed the imaging visits, the Data Monitoring Committee will review the images. The visual assessment of the scans in these first 20 participants will support the continuation or the termination of the Phase II study.



Version: 01 Page: **21 of 167** 

The following table summarizes all the procedures and evaluations to be conducted during the study:

| Study Procedures | Screening<br>(Within 8<br>weeks prior<br>to Day 0) | SPECT/CT<br>Visit<br>(Day 0) | 24 hours<br>post IP<br>injection <sup>1</sup> | 30 ± 3 days<br>post IP<br>injection<br>(Day 30) |
|---|---|---|---|---|
| Written informed consent | X | | | |
| Inclusion/exclusion criteria | X | X | | |
| Medical history | Х | | | |
| Concomitant medications | Х | X | Χ | X |
| Physical examination (height, weight, BMI) | Х | х | | |
| Vital signs<br>(BP, HR) | × | × | | |
| Lab analysis (hematology, PT/PTT/INR, biochemistry, urine) | × | | | Х |
| Immunogenicity by ELISA <sup>2</sup> | Х | | | Х |
| Pregnancy test | Х | X | | |
| Carotid ultrasound <sup>3</sup> | Х | | | |
| rh-Annexin V-128 administration | | Х | | |
| Planar & SPECT/CT imaging | | Х | | |
| Adverse events assessment | | Х | Х | Х |

<sup>&</sup>lt;sup>1</sup>Within 24 hours after injection of <sup>99m</sup>Tc-rhAnnexin V-128, each participant will be called to review any signs or symptoms of AEs.

#### 4.3.5 Planned sample size

The primary hypothesis is that <sup>99m</sup>Tc-rhAnnexin V-128 carotid imaging can detect apoptosis. We anticipate that the prevalence of positive <sup>99m</sup>Tc-rhAnnexin V-128 carotid scans will be about 0.3 to 0.5 of the patients. A sample size of 30 patients produces a 95% confidence interval with a precision of about 0.17 to 0.20 when the estimated proportion is 0.3 to 0.5. Sample size was also estimated for the comparison of <sup>99m</sup>Tc-rhAnnexin V-128 uptake in asymptomatic or symptomatic with TIA patients with carotid disease versus normals using a 5% significance level and power of 95%. The measured neck uptake in 12 normals was 0.8 ± 0.27% ID/gm in the Phase I study. Assuming a similar SD of 0.27% ID/gm in the patients and a minimal clinically important difference (MCID) of

<sup>&</sup>lt;sup>2</sup>Anti-rhAnnexin V-128 IgG and IgM antibodies will be quantified in serum samples by ELISA. For this purpose 10 mL blood samples will be collected at screening and Day 30 (±3 days) post administration of investigation product. Serum will be prepared, divided into six aliquots and frozen (-80°C). Three out of six serum samples per time-point will then be shipped to the central laboratory.

<sup>&</sup>lt;sup>3</sup>Within 8 weeks prior to <sup>99m</sup>Tc-rhAnnexin V-128 SPECT imaging.





Version: 01 Page: **22 of 167** 

50% or a change of 0.4 in uptake, the required sample size is 9 normals and 25 patients. Allowing for attrition, we plan to recruit 10 normals and 35 patients.





## 5 SUBJECT POPULATIONS (ANALYSIS SETS)

## 5.1 Efficacy

#### 5.1.1 Full analysis set (FAS)

In accordance with the Intention To Treat (ITT) principle, the FAS population includes all subjects who received the study drug and completed the <sup>99m</sup>Tc-rhAnnexin V-128 imaging procedure.

#### 5.1.2 Per Protocol population (PP)

All subjects in the FAS population for whom no major protocol violations/deviations occurred. The criteria defining the major protocol deviations will be established before the data base locking.

## 5.2 Safety set

The safety population is made up of all subjects who received the administration of <sup>99m</sup>Tc-rhAnnexin V-128.

## 5.3 Primary population

The primary and secondary efficacy analysis will be based on the FAS population.

The primary efficacy analysis on the Primary endpoint of Phase II will be also performed on the PP population as supportive analysis.

The assessment of safety and tolerability will be based on the Safety population.



Version: 01 Page: **24 of 167** 

#### 6 STATISTICAL METHODS

### 6.1 Statistical analysis strategy

The statistical analyses will be performed in accordance with the principles of ICH E9 guideline and the guideline on clinical evaluation of diagnostic agents and they will be based on data from the study site, unless otherwise stated.

The statistical analysis will be performed by \_\_\_\_\_\_ - Italy

#### 6.1.1 General statistical considerations

For continuous variables, descriptive summary statistics will include the number of non-missing values, number of missing values, mean, standard deviation, 95% 2-sided confidence interval, median, lower and upper quartile, minimum and maximum. Box plot graphs will also be presented when appropriate.

For categorical variables, descriptive summary statistics will include counts and percentages per category.

For analysis purposes, baseline for a given assessment will be defined as the last non-missing value prior to the administration of <sup>99m</sup>Tc-rhAnnexin V-128, unless stated otherwise.

#### 6.1.2 Efficacy endpoint(s)

#### 6.1.2.1 Primary endpoint of PoC

The feasibility of imaging apoptotic activity in carotid atherosclerotic plaques using <sup>99m</sup>Tc-rhAnnexin V-128 will be assessed by the data monitoring committee (visual image review and consensus) using the first 15 patient and 5 control scans.

The frequency and severity of abnormal carotid scans will be determined in the patient and control groups by review of the number, localization, length and uptake intensity grade of each plaque to define a positive or negative scan at each time point.

DMC outputs were defined in the DMC charter.





#### 6.1.2.2 Primary endpoint of Phase II

The primary endpoint of Phase II is the prevalence of abnormal <sup>99m</sup>Tc-rhAnnexin V-128 Planar and SPECT/CT scans in patient and control groups.

The prevalence of apoptotic activity is defined as the proportion of patients with "abnormal" SPECT imaging scans (also described as positive scans). Activity concentrations (MBq/cc or % injected dose/gram) determined from reconstructed image counts as described in section 4.3.3.3 will be compared with the normal database of carotid and aortic uptake from the 10 control participants and used to identify abnormal uptake in carotid artery disease participants that will define an abnormal SPECT/CT result.

The prevalence of abnormal <sup>99m</sup>Tc-rhAnnexin V-128 scans will be reported with the related 95% C.I. for both carotid participating group and the control group at each time point and overall.

The overall result of <sup>99m</sup>Tc-rhAnnexin V-128 imaging will be unique: patients with at least one SPECT/CT positive result (after 60 min or after 120 min from <sup>99m</sup>Tc-rhAnnexin V-128 injection) will be considered as abnormal, patients with both SPECT/CT images negative will be considered as normal.

The results of <sup>99m</sup>Tc-rhAnnexin V-128 will also be reported in contingency tables as normal and abnormal for each group (patient and control) at each time point (60 min and 120 min after injection) in order to assess where any difference between the time points occurred.

Results of Carotid Ultrasound and SPECT procedures will be included in the data listing. The listings will also flag which patients had a history of TIA.

The primary efficacy analysis will be performed on the FAS population.

#### 6.1.2.3 Secondary endpoints

The secondary endpoints of Phase II and the related statistical analysis are:

- Descriptive statistics of <sup>99m</sup>Tc-rhAnnexin V-128 uptake in patients vs control participants will be presented by areas of interest (left carotid, right carotid, thoracic aorta, abdominal aorta and aortic arch) and by time points to assess the background uptake profile and the pathologic profile. Comparison of uptake in patients vs controls at each timepoint will be explored by the most appropriate test i.e. two sample t-test.
- The relationship between carotid uptake (separately for left and right) and ultrasound grade of plaque echolucency/echogenicity (1 echolucent, 2 predominantly echolucent, 3 predominantly echogenic, 4 echogenic) will be assessed for all patients using box plots and



Version: 01 Page: **26 of 167** 

summaries of uptakes by the levels of echolucency/echogenicity for each time point. Only carotids with stenosis (defined as  $\geq$  50% as per protocol) will be included in this analysis (i.e. a patient with only 1 carotid with stenosis  $\geq$  50% will contribute data for that carotid uptake value and the associated plaque echolucency/echogenicity value for the same carotid, patients with stenosis in both carotids will contribute data on uptake and echolucency/echogenicity for each of their carotids).

Association between carotid and aortic uptake will be assessed for patients and controls, by time
point, using scatter plots. All carotids with ≥ 50% stenosis (as described above) will be included
in this plot, and different colours/symbols will be used for left and right carotid results. If further
investigation is considered appropriate, the correlation coefficients (Pearson's or Spearman's)
within left carotids and right carotids separately will be calculated.

#### 6.1.3 Safety endpoint(s)

Safety and tolerability will be primarily evaluated by the incidence of adverse events, clinical laboratory values (hematology, blood chemistry and urinalysis), development of anti-Annexin V-128 antibodies, vital signs (blood pressure and heart rate) and physical examination findings.

All safety data will be included in the data listings and summary tables will be based on the safety population. The statistical analysis of safety data will be mainly descriptive in nature.

#### 6.1.3.1 Adverse events

All original AE/SAE terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 19.0.

Adverse events (AEs) will be listed on an individual basis, including relationship and severity, LLT (Lowest Level Term) and verbatim term. Treatment emergent Adverse events (TEAEs) and Adverse Drug Reactions (ADRs) will be summarized by System Organ Class (SOC) and Preferred Term (PT), grouping patients versus control subjects, and also including a total column for all subjects who received Annexin. Participants with more than one adverse event within a particular SOC and PT will be counted only once for that SOC and PT reporting the highest level in severity. The incidence of TEAEs and ADRs will also be summarized by subject type and severity.

Listings and summaries of serious adverse events (SAEs), adverse events leading to withdrawal and listings of deaths will also be presented.

Treatment Emergent Adverse Events and Adverse Drug Reactions will be defined as below:



Version: 01 Page: **27 of 167** 

- Treatment Emergent Adverse Events: Events that emerge after the <sup>99m</sup>Tc-rhAnnexin V-128 injection and up to 30 days after the injection that were absent before it or worsen relative to the pre-treatment state.
- Adverse Drug Reactions: Treatment emergent adverse events possibly or probably related to study treatment.

#### 6.1.3.2 Clinical laboratory values

Hematology, blood chemistry, urinalysis and immunogenicity values are recorded at baseline for screening,  $30 \pm 3$  days post IP administration and following any adverse events. Descriptive statistics including shift tables will be generated for all laboratory tests performed i.e. the actual values and the changes from pre-injection.

Data listing will be ordered by subject and measuring time. Listings of abnormal results (both clinically and non-clinically relevant) will also be reported.

#### 6.1.3.3 Vital signs and physical examination

Vital signs and physical examination data are recorded once at screening visit and twice at imaging visit (SPECT/CT Visit, Day 0), before the injection of <sup>99m</sup>Tc-rhAnnexin V-128 and at the end of SPECT/CT (after the <sup>99m</sup>Tc-rhAnnexin V-128 injection). Descriptive statistics will be tabulated by measuring time for raw data and changes from baseline. Data listings will be ordered by subject and measuring time.

#### 6.1.4 Missing data and outliers

#### 6.1.4.1 Missing data

As stated in the protocol, missing data will not be replaced.

#### 6.1.4.2 Missing or incomplete dates

Incomplete dates due to missing day will be recorded as full dates replacing the missing day with the first day of month (01). Incomplete dates due to missing day and month will be recorded as full dates replacing the missing day and month with the first day of month and first month of the year (01/January). The trial database will record the information about incomplete dates due to missing day or due to missing day and month.



Version: 01 Page: **28 of 167** 

Only the incomplete dates related to medical history (date of diagnosis and end date), concomitant medications (start and end date) and AEs (start and end date) will be replaced according to the above rule.

Calculation, sorting or assignation based on dates, in case of incomplete dates, will be performed using the related full dates defined by the above rule.

In all listings, missing dates will be missing and incomplete dates will be reported as full dates. In all listings will also be reported the information about incomplete dates according to the following coding: missing value = full date, Day = missing day, Day&Month = missing day and month.

#### 6.1.4.3 **Outliers**

For categorical or score data, like adverse events, physical exam's findings and disease assessment parameters, outliers are not expected.

Demographic, vital signs, and clinical laboratory (hematology, blood chemistry and urinalysis) parameters will be checked for outliers according to data plausibility, normal ranges and the range between mean  $\pm 2$  S.D.

For each identified outlier, will inform the Sponsor in order to assess any errors. If data cannot be verified or if relevant, the descriptive statistics of the related parameters will be reported with and without the outliers. If appropriate, outliers can also be specifically identified in the boxplots.

#### 6.1.5 Subject disposition

A listing of dates of assessments (relative day) and their study exposure will be presented by subject.

A summary table and a flow chart will be presented for each subject population presenting the number of subjects at each assessment procedure and identifying the number of subjects who withdrew over time.

#### 6.1.6 Withdrawals

Discontinued subjects will be listed and a summary table of the number and percentage of subjects who withdrew from the study and the reasons for withdrawal will be presented for all screened subjects.



Version: 01 Page: **29 of 167** 

#### 6.1.7 Demographic and baseline characteristics

All demographic and baseline characteristics will be listed by subject. Summary statistics will be provided for demographic and baseline characteristics for FAS and Safety population (if different from FAS).

#### 6.1.8 Medical and surgical history

Medical and surgical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 19.0.

Medical and surgical history will be listed on an individual basis, including Preferred Term (PT) and verbatim term; the listings will be sorted by subject.

A frequency table of the number and percentage of subjects will be provided for all medical and surgical history by primary SOC and PT for Safety population.

#### 6.1.9 Subject compliance

After reconstitution and radiolabeling, <sup>99m</sup>Tc-rhAnnexin V-128 is administered as a single intravenous bolus of 350 MBq ± 10% at the imaging visit (Day 0). The administered dose recorded in the eCRF will not be the difference between the pre-injection dose and the post-injection residual dose but will be the decay corrected dose which takes into account the natural product half-life.

A listing will be presented for imaging product administration (dose, quality, date) by subject. Deviations from observed and scheduled times will be presented. Summary tables will be presented for all the continuous variables.

A listing will be presented for concomitant medications.

All the protocol deviations will be also listed by subject.

#### 6.1.10 Prior and concomitant medications

Concomitant medications will be coded using ATC Drug Dictionary Version 2016.

Listings will be presented for ATC name (third level) and verbatim text. The listings will be sorted by subject, chronological start date, ATC name, verbatim text and active substance.

A frequency table of the number and percentage of subjects will be provided for concomitant medications by pharmacological subgroup and chemical substance for Safety population. Two different tables will report Prior Medications (the medications taken and stopped within 30 days prior the <sup>99m</sup>Tc-rhAnnexin V-128 injection) and Prior and Concomitant Medications (the medications



Version: 01 Page: **30 of 167** 

started within 30 days prior the <sup>99m</sup>Tc-rhAnnexin V-128 injection and continued after the <sup>99m</sup>Tc-rhAnnexin V-128 injection and the medications started after the <sup>99m</sup>Tc-rhAnnexin V-128 injection).

#### 6.1.11 Derived data

The derived data are variables which are calculated from the raw data in the CRF and not included in the database (e.g.: Age, BMI). The formula used for derived data and the strategy for missing data are provided in Section 12.1.

#### 6.1.12 Visit windows

The screening visit can occur anytime within 8 weeks before the injection day (Day 0).

The first follow-up visit (phone call) should occur within 24 hours after the injection. The second follow-up visit should occur 30 days after the injection with a window of 3 days, i.e. the visit has to be performed between the 27<sup>th</sup> and the 33<sup>rd</sup> day from the <sup>99m</sup>Tc-rhAnnexin V-128 administration.

#### 6.1.13 Rules and data formats

Data will be presented using an appropriate number of decimal places (i.e. the number of decimal places used does not imply undue precision). Raw data will be presented to the number of decimal places collected, and derived data will be presented to an appropriate number of decimal places. The appropriate number of decimal places will be determined by general practice, mathematical rationale or scientific rationale (e.g. age should be presented in whole numbers).

For summary statistics, the following will be presented: number of non-missing values (n), number of missing values, arithmetic mean, standard deviation, median, the IQR (first quartile, third quartile), the range (minimum, maximum) and, only if appropriate, 95% 2-sided confidence interval.

Mean, standard deviation, first quartile, median, third quartile and confidence interval values will be rounded to one more decimal place than the raw data whereas minimum and maximum will be reported with the same precision as the raw data.

Percentages will be reported to one decimal place. Percentages will be calculated using a denominator of all subjects in a specified population. The denominator will be specified in a footnote to the tables for clarification if necessary.

p-values will be reported to four decimal places (e.g., p=0.0037), after rounding; p-values which are less than 0.0001 will be presented as "<0.0001".



Version: 01 Page: **31 of 167** 

All text fields must be left justified and numeric or numeric with some text specification (e.g., not done, unknown, <4.5, ...) must be decimal justified. Dates will be presented in the format [dd/mm/yyyy] and times in the format [hh:mm] using 24-hour clock scale.

#### 6.1.14 Pooling of centres

Not applicable.

#### 6.1.15 Interim analysis

No formal interim analysis will be done; however the DMC will analyse Planar and SPECT/CT images of the first 15 patients and of the first 5 controls in order to determine the feasibility of imaging apoptotic activity in carotid atherosclerotic plaques of asymptomatic or symptomatic with TIA patients with significant carotid disease, by using <sup>99m</sup>Tc-rhAnnexin V-128 imaging, and to report the prevalence of abnormal <sup>99m</sup>Tc-rhAnnexin V-128 scans.

## 6.1.16 Role of independent data monitoring committee (DMC) / interim data review committee

The Data Monitoring Committee (DMC) consists of investigators and Sponsor representatives, as well as external persons such as independent experts, if deemed necessary by the Sponsor. The main function of the committee will be to review and evaluate the images of the first 15 patients and of the first 5 healthy participants in terms of image quality, carotid target uptake and clinical relevance of the study product. The DMC will also review the safety data. The frequency of abnormal carotid scans will be determined in the participant and control groups. The study will be terminated if there is a low frequency of positive scans in the carotid participant group or high frequency of positive scans in the control group.

The DMC will promptly give recommendations to continue or terminate the study. The DMC report will be prepared by the Sponsor and sent to the REB and regulatory authorities as required. Preliminary results can be used by the Sponsor for publication purpose, before the end of the main trial.

#### 6.1.17 Covariates and analysis of subgroups

The analysis on the efficacy endpoints will be performed on the two groups of enrolled subjects (patients and control group). Patient group will also be divided into two groups (normal and abnormal) depending on imaging results (negative or positive).




Version: 01 Page: **32 of 167** 

If deemed relevant some additional analysis might be conducted to explore the impact of clinically relevant covariates such as the level of carotid stenosis (as determined by ultrasound), history of TIA and any other relevant factors on the results.

#### 6.1.18 Sensitivity analysis

Not Applicable.

## 6.1.19 Multiplicity

As stated in the protocol, no adjustments will be made for multiplicity.

## 6.1.20 Significance testing and estimation

All statistical tests will be two-sided at the 5% level of significance.





## 7 COMPUTER SYSTEMS, SOFTWARE AND VALIDATION OF PROGRAMS

#### 7.1 Hardware

The statistical analysis will be performed using Dell personal computer with Windows 7 professional (64 bit) as operating system.

#### 7.2 Software

All tables, listings and figures will be produced and statistical analysis performed using SAS version 9.4. All output will be in Word format.

### 7.3 Validation programs

An Independent Statistician is responsible for reviewing each project program and output associated with the deliverable product. Program logs are reviewed for logical, syntax and fatal errors. The review in SAS includes, but is not limited to, all ERRORS, WARNINGS, NOTES, and variables check. Program logs are also reviewed for accurate and consistent variable and observation counts following each procedure and data step.

The Independent Statistician is also responsible for checking and reviewing the work produced using whatever method he/she feels is appropriate (e.g. SAS commands review, hand calculation, etc.) to reassure of the quality of the output.

Outputs are reviewed for typographical errors, misspellings and nonsensical values or results and to check the consistency with the reporting and analysis plan. Outputs are cross-checked against each other for accuracy and consistency. For statistical tables, listings, and figures, this procedure includes comparison of subject group numbers, counts of subjects at each observation point, and consistency of results for variables between outputs.

Findings of the quality control reviews are communicated to the party responsible for making necessary changes. The programs will be retested after modifications.

After final review, and when no further changes are required to produce the deliverables, the Independent Statistician needs to complete and sign the SAS Outputs, to indicate that he has successfully performed all of his responsibilities.




Version: 01 Page: **34 of 167** 

## **8 CHANGES FROM PROTOCOL**

No changes from the protocol were made.

# Statistical Analysis Plan ANNEXIN 04 Confidential

Version: 01

Page: **35 of 167** 

## 9 REFERENCES

Not applicable.



Version: 01 Page: **36 of 167** 

#### **10 DATA PRESENTATION**

Data listings are presented for all screened subjects.

Footnotes should be used to clarify ambiguities (e.g.: the denominator used to calculate a percentage or notes for the programmer). If the number of footnotes is high, they could be presented only in the last page, with on each page the following footnote "See last page for listing notes". The order of the footnotes for key symbols (\*, ~) will be in the order that they appear in the listing.

### 10.1 Listings index

#### **16.2 SUBJECT DATA LISTINGS**

#### 16.2.1 Discontinued subjects

Listing 16.2.1.1: Subject Disposition – All Subjects

Listing 16.2.1.2: Subject Disposition – Study Withdrawals

Listing 16.2.1.3: Inclusion Criteria

Listing 16.2.1.4: Exclusion Criteria

Listing 16.2.1.5: Screening Failures

#### 16.2.2 Protocol deviations

Listing 16.2.2: Protocol Deviations and Reasons for Exclusion from the Study

**Populations** 

#### 16.2.3 Subjects excluded from the efficacy analysis

Not applicable

#### 16.2.4 Demographic data

Listing 16.2.4.1: Demographics

Listing 16.2.4.2: Carotid Ultrasound

Listing 16.2.4.3: Medical History and Associated Pathologies

Listing 16.2.4.4: Prior and Concomitant Medications

#### 16.2.5 Compliance and/or drug concentration data

Listing 16.2.5.1: Study Drug Administration and Extent of Subject Exposure

#### 16.2.6 Individual efficacy response data

Listing 16.2.6.1: Carotid and Aorta Imaging Assessment

Version: 01 Page: **37 of 167** 

Listing 16.2.6.2: Carotid and Aorta Imaging Assessment – Uptake – Data Recorded

on DMC Assessement Form

### 16.2.7 Adverse event listings (each subject)

Listing 16.2.7.1: All Adverse Events

Listing 16.2.7.2: Serious Adverse Events

Listing 16.2.7.3: Adverse Events Leading to Withdrawal

Listing 16.2.7.4: Adverse Events with Outcome Death

#### 16.2.8 Listing of individual laboratory measurements by subject

Listing 16.2.8.1: Hematology

Listing 16.2.8.2: Blood Chemistry

Listing 16.2.8.3: Urinalysis

Listing 16.2.8.4: Immunogenicity

### 16.2.9 Listing of other safety data

Listing 16.2.9.1: Pregnancy Test

Listing 16.2.9.2: Physical Examination

Listing 16.2.9.3: Vital Signs

### 10.2 Listing templates

Listing templates are provided in Appendix 11.1. The listings will be presented in landscape, in a fixed font (Arial) with a minimum size as 8.

### 10.3 Tables index

#### 14. TABLES, FIGURES AND GRAPHS

#### 14.1 DEMOGRAPHIC DATA

Table 14.1.1: Subject Disposition

Table 14.1.2: Analysis Populations

Table 14.1.3: Protocol Deviations

Table 14.1.4.1: Demographics – FAS Population

Table 14.1.5.1: Carotid Ultrasound – FAS Population

### Confidential

Page: **38 of 167** 

| Table | 14.1.6.1: | Medical History and Associated Pathologies – Safety Population |
|---|---|---|
| Table | 14.1.7.1: | Prior Medications or Non-Drug Tharapies – Safety Population |
| Table | 14.1.7.2: | Prior and Concomitant Medications or Non-Drug Therapies – Safety Population |
| Table | 14.1.8.1: | Study Drug Administration – Safety Population |
| 14.2 EFFICACY | DATA | |
| Table | 14.2.1.1: | Carotid and Aorta Imaging Assessment – Prevalence of Positive Scans – FAS Population |
| Table | 14.2.1.2: | Carotid and Aorta Imaging Assessment – Prevalence of Positive Scans – PP Population |
| Table | 14.2.1.3: | Patient Carotid and Aorta Imaging Assessment – Comparison between time point – FAS Population |
| Table | 14.2.1.4: | Left Carotid Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population |
| Table | 14.2.1.5: | Right Carotid Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population |
| Table | 14.2.1.6: | Thoracic Aorta Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population |
| Table | 14.2.1.7: | Abdominal Aorta Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population |
| Table | 14.2.1.8: | Aortic Arch Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population |
| Table | 14.2.1.9: | Left Carotid Uptake Imaging Assessment by ultrasound grade of plaque echolucency/echogenicity – Target to Background Ratio (TBR) – Patients - FAS Population |
| Table | 14.2.1.10: | Right Carotid Uptake Imaging Assessment by ultrasound grade of plaque echolucency/echogenicity – Target to Background Ratio (TBR) – Patients - FAS Population |

Version: 01

### **14.3 SAFETY DATA**

## 14.3.1 Displays of Adverse Events

Table 14.3.1.1: Overall Summary of Adverse Events – Safety Population


| Table 14.3.1.2: | Number (%) of Subjects Reporting Treatment Emergent Adverse |
|---|---|
| | Events by Primary System Organ Class and Preferred Term - |
| | Safety Population |
| Table 14.3.1.3: | Number (%) of Subjects Reporting Treatment Emergent Adverse |
| | Events by Severity – Safety Population |
| Table 14.3.1.4: | Number (%) of Subjects Reporting Adverse Drug Reactions by |
| | Severity – Safety Population |
| Table 14.3.1.5: | Number (%) of Subjects Reporting Treatment Emergent Serious |
| | Adverse Events by Primary System Organ Class and Preferred |
| | Term – Safety Population |
| Table 14.3.1.6: | Number (%) of Subjects Reporting Treatment Emergent Serious |
| | Adverse Events by Severity – Safety Population |
| Table 14.3.1.7: | Number (%) of Subjects Reporting Serious Adverse Drug Reactions |
| | by Severity – Safety Population |

### 14.3.2 Listings of Deaths, Other Serious and Significant Adverse Events

Version: 01

Table 14.3.2.1: Listing of Adverse Events with Outcome Death – Safety Population

Table 14.3.2.2: Listing of Serious Adverse Events – Safety Population

#### 14.3.3 Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events

Only raw narratives will be presented in this section if any.

#### 14.3.4 Abnormal Laboratory Value Listing (each patient)

Only patients with clinically significant abnormal laboratory value(s) will be presented in this section if any.

Table 14.3.4: Abnormal Laboratory Value Listing (Each Patient) – Safety Population

### 14.3.5 Laboratory Measurements

Table 14.3.5.1: Hematology – Safety Population

Table 14.3.5.2: Blood Chemistry – Safety Population

Table 14.3.5.3: Urinalysis – Safety Population

#### 14.3.6 Other Safety Data

Table 14.3.6.1: Vital Signs – Safety Population



Version: 01 Page: **40 of 167** 

## 10.4 Table templates

Table templates are provided for each unique table in Appendix 11.2. The tables will be presented in landscape, in a fixed font (arial) with a minimum size as 8.

All tables, in table number order, must be presented in a single Word file.

# 10.5 Figures index

### 14. TABLES, FIGURES AND GRAPHS

### **14.2 EFFICACY DATA**

| Figure 14.2.1.1: | Left Carotid Target to Background Ratio (TBR) Imaging Assessment - Patients – Carotid with Stenosis ≥ 50% – FAS Population - 60 mins after IP injection |
|---|---|
| Figure 14.2.1.2: | Left Carotid Target to Background Ratio (TBR) Imaging Assessment - Patients – Carotid with Stenosis ≥ 50% – FAS Population - 120 mins after IP injection |
| Figure 14.2.1.3: | Right Carotid Target to Background Ratio (TBR) Imaging Assessment - Patients - Carotid with Stenosis ≥ 50% - FAS Population 60 mins after IP injection |
| Figure 14.2.1.4: | Right Carotid Target to Background Ratio (TBR) Imaging Assessment - Patients - Carotid with Stenosis ≥ 50% - FAS Population - 120 mins after IP injection |
| Figure 14.2.1.5: | Scatterplot between Left and Right Carotid and Thoracic Aorta Target to Background Ratio (TBR) – Patients – FAS Population - 60 mins after IP injection |
| Figure 14.2.1.6: | Scatterplot between Left and Right Carotid and Thoracic Aorta Target to Background Ratio (TBR) – Patients – FAS Population - 120 mins after IP injection |
| Figure 14.2.1.7: | Scatterplot between Left and Right Carotid and Abdominal Aorta Target to Background Ratio (TBR) – Patients – FAS Population - 60 mins after IP injection |




| Figure 14.2.1.8: | Scatterplot between Left and Right Carotid and Abdominal Aorta |
|---|---|
| | Target to Background Ratio (TBR) - Patients - FAS Population - |
| | 120 mins after IP injection |
| Figure 14.2.1.9: | Scatterplot between Left and Right Carotid and Aortic Arch Target |
| | to Background Ratio (TBR) – Patients – FAS Population - 60 mins |
| | after IP injection |
| Figure 14.2.1.10: | Scatterplot between Left and Right Carotid and Aortic Arch Target |
| | to Background Ratio (TBR) – Patients – FAS Population - 120 mins |

## 10.6 Figure templates

Figure templates are provided for each unique figure in Appendix 11.3. The figures will be presented in landscape, in a fixed font (arial) with a minimum size as 8.

All figures, in figure number order, must be presented in a single Word file.

after IP injection

Version: 01

## 10.7 Statistical appendix

A statistical appendix for inclusion in the study report will be provided. All the methods used in checking the assumptions of the analyses and conclusions should be included and explained. Transformation of the data or other methods used for the statistical analysis other than the ones detailed in the SAP will be described and the change will be justified. All the SAS output will be included without reworking the data (raw output).

This output should contain the study number, the date, the number of pages printed by SAS and the table number to which it refers. Any other relevant information (e.g. statistical references...) will be added in the statistical appendix.



Version: 01 Page: **42 of 167** 

### 11 APPENDICES

# 11.1 Standard listings

All listings must contain examples of possible data and be presented in fixed font (arial) with a minimum size as 8.





Version: 01 Page: **43 of 167** 

## **Listing 16.2.1.1:** Subject Disposition – All Subjects

| Subject ID | Screening date | Informed consent date | Subject group* | Visit 1 date | Phone call 2 date | Visit 3 date | Premature study discontinuation date | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_FIRSTVISITDAT<br>E | PAT_INFCONS_DATE | PAT_INFCONS_TYPE | PATV_VISITDATE | PATV_VISITDATE | PATV_VISITDATE | SD_DATE | [Derived data] | [Derived data] | [Derived data] |
| 04-CA-001 | 11/03/2011 | 11/03/2011 | Patient | 11/04/2011 | 12/04/2011 | 11/05/2011 | | Yes | Yes | Yes |
| 04-CA-002 | 09/04/2011 | 09/04/2011 | Control | 09/04/2011 | 10/04/2011 | 10/05/2011 | | Yes | Yes | Yes |
| 04-CA-003 | 10/07/2011 | 10/07/2011 | Control | 15/07/2011 | 16/07/2011 | NA | 10/08/2011 | Yes | No | Yes |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_SD.

Note: NA = Not Available for patient early withdrawal

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **44 of 167** 

### Listing 16.2.1.2: Subject Disposition – Study Withdrawals

| Subject ID | Screening date | Informed consent date | Informed consent type* | Premature study discontinuation date | Reason for withdrawal | Explanation | Notes | FAS | PP | Safety | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_FIRSTVISITDATE | PAT_INFCONS_DATE | PAT_INFCONS_TYPE | SD_DATE | SD_OUTCOME | SD_OUTCOME_SP | SD_NOTES | [Derived data] | [Derived data] | [Derived data] | |
| 04-CA-001 | 11/03/2011 | 11/03/2011 | Patient | 10/05/2012 | XXXXXX | XXXXXX | XXXXXX | Yes | No | Yes | |
| 04-CA-002 | 09/04/2011 | 09/04/2011 | Control | 10/05/2012 | XXXXXX | XXXXXX | XXXXXX | Yes | No | Yes | |
| 04-CA-003 | 10/07/2011 | 10/07/2011 | Control | 10/05/2012 | XXXXXX | XXXXXX | XXXXXX | Yes | No | Yes | |
| | PAT_PATNUMBER 04-CA-001 04-CA-002 | PAT_PATNUMBER PAT_FIRSTVISITDATE 04-CA-001 11/03/2011 04-CA-002 09/04/2011 | PAT_PATNUMBER PAT_FIRSTVISITDATE PAT_INFCONS_DATE 04-CA-001 11/03/2011 11/03/2011 04-CA-002 09/04/2011 09/04/2011 | PAT_PATNUMBER PAT_FIRSTVISITDATE PAT_INFCONS_DATE PAT_INFCONS_TYPE 04-CA-001 11/03/2011 11/03/2011 Patient 04-CA-002 09/04/2011 09/04/2011 Control | Subject IDScreening dateInformed consent dateInformed consent type*discontinuation datePAT_PATNUMBERPAT_FIRSTVISITDATEPAT_INFCONS_DATEPAT_INFCONS_TYPESD_DATE04-CA-00111/03/201111/03/2011Patient10/05/201204-CA-00209/04/201109/04/2011Control10/05/2012 | Subject IDScreening dateInformed consent dateInformed consent type*discontinuation datewithdrawalPAT_PATNUMBERPAT_FIRSTVISITDATEPAT_INFCONS_DATEPAT_INFCONS_TYPESD_DATESD_OUTCOME04-CA-00111/03/201111/03/2011Patient10/05/2012XXXXXXX04-CA-00209/04/201109/04/2011Control10/05/2012XXXXXXX | Subject IDScreening dateInformed consent dateInformed consent type*discontinuation datewithdrawalExplanationPAT_PATNUMBERPAT_FIRSTVISITDATEPAT_INFCONS_DATEPAT_INFCONS_TYPESD_DATESD_OUTCOMESD_OUTCOME_SP04-CA-00111/03/201111/03/2011Patient10/05/2012XXXXXXXXXXXXX04-CA-00209/04/201109/04/2011Control10/05/2012XXXXXXXXXXXXXX | Subject IDScreening dateInformed consent dateInformed consent type*discontinuation datewithdrawalExplanationNotesPAT_PATNUMBERPAT_FIRSTVISITDATEPAT_INFCONS_DATEPAT_INFCONS_TYPESD_DATESD_OUTCOME_SPSD_NOTES04-CA-00111/03/201111/03/2011Patient10/05/2012XXXXXXXXXXXXXXXXXXXXX04-CA-00209/04/201109/04/2011Control10/05/2012XXXXXXXXXXXXXXXXXXXXX | Subject IDScreening dateInformed consent dateInformed consent type*discontinuation datewithdrawalExplanationNotesFASPAT_PATNUMBERPAT_FIRSTVISITDATEPAT_INFCONS_DATEPAT_INFCONS_TYPESD_DATESD_OUTCOME_SPSD_NOTES[Derived data]04-CA-00111/03/201111/03/2011Patient10/05/2012XXXXXXXXXXXXXXXXXXXXXYes04-CA-00209/04/201109/04/2011Control10/05/2012XXXXXXXXXXXXXXXXXXXXXYes | Subject IDScreening dateInformed consent dateInformed consent type*discontinuation datewithdrawalExplanationNotesFASPPPAT_PATNUMBERPAT_FIRSTVISITDATEPAT_INFCONS_DATEPAT_INFCONS_TYPESD_DATESD_OUTCOME_SPSD_NOTES[Derived data]04-CA-00111/03/201111/03/2011Patient10/05/2012XXXXXXXXXXXXXXXXXXXXXYesNo04-CA-00209/04/201109/04/2011Control10/05/2012XXXXXXXXXXXXXXXXXXXXXYesNo | Subject IDScreening dateInformed consent dateInformed consent type*discontinuation datewithdrawalExplanationNotesFASPPSafetyPAT_PATNUMBERPAT_FIRSTVISITDATEPAT_INFCONS_DATESD_DATESD_OUTCOMESD_OUTCOME_SPSD_NOTES[Derived data][Derived data]04-CA-00111/03/201111/03/2011Patient10/05/2012XXXXXXXXXXXXXXXXXXXXXYesNoYes04-CA-00209/04/201109/04/2011Control10/05/2012XXXXXXXXXXXXXXXXXXXXXYesNoYes |

Data Source Table: W\_PATIENT, W\_SD.

Note: NA = Not Available for patient early withdrawal

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **45 of 167** 

### Listing 16.2.1.3: Inclusion Criteria

| | | | | | | | Inclusion criteri | а | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Sex | Age | Screening date | First | Second | Third | Fourth | Fifth |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | PAT_GENDER | PAT_AGEYEAR | PAT_FIRSTVISITDATE | IC_1 | IC_2 | IC_3 | IC_4 | IC_5 |
| 04-CA-001 | Patient | Male | 54 | 11/03/2011 | Yes | Yes | Not applicable | Yes | Yes |
| 04-CA-002 | Control | Female | 68 | 09/04/2011 | Yes | Yes | Yes | Not applicable | Not applicable |
| 04-CA-003 | Control | Female | 59 | 10/07/2011 | No | Yes | Yes | Yes | No |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IEC.

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 

## Listing 16.2.1.4: Exclusion Criteria

| Exclusio | n criteria | | | |
|----------|------------|-------|---------|--------|
| Fourth | Fifth | Sixth | Seventh | Eighth |
| EC_4 | EC_5 | EC_6 | EC_7 | EC_8 |

| Subject ID | Subject group* | Sex | Age | Screening date | First | Second | Third | Fourth | Fifth | Sixth | Seventh | Eighth |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS<br>_TYPE | PAT_GENDER | PAT_AGEYEA<br>R | PAT_FIRSTVISITDATE | EC_1 | EC_2 | EC_3 | EC_4 | EC_5 | EC_6 | EC_7 | EC_8 |
| 04-CA-001 | Patient | Male | 54 | 11/03/2011 | No | No | Not applicable | No | No | No | No | No |
| 04-CA-002 | Control | Female | 68 | 09/04/2011 | No | Yes | No | No | No | No | No | No |
| 04-CA-003 | Control | Female | 59 | 10/07/2011 | Yes | No | No | No | No | No | No | No |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IEC.

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **47 of 167** 

## Listing 16.2.1.5: Screening Failures

| Subject ID | Subject group* | Screening failure | Reason for screen failure |
|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | [Derived data] | [Derived data] |
| 04-CA-001 | Patient | Yes | XXXXX |
| 04-CA-002 | Control | No | XXXXX |
| 04-CA-003 | Control | No | XXXXX |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IEC, W\_SD.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **48 of 167** 

### Listing 16.2.2: Protocol Deviations and Reasons for Exclusion from the Study Populations

| Subject ID | Subject group* | Screening date | FAS | PP | Safety | Deviation description | Reason for exclusion |
|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | PAT_FIRSTVISITDATE | [Derived data] | [Derived data] | [Derived data] | [Derived data] | [Derived data] |
| 04-CA-001 | Patient | 11/03/2011 | Yes | Yes | No | XXXXXX | XXXXXX |
| 04-CA-002 | Control | 09/04/2011 | No | Yes | Yes | XXXXXX | XXXXXX |
| 04-CA-003 | Control | 10/07/2011 | Yes | No | Yes | XXXXXX | XXXXXX |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_SD.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **49 of 167** 

## **Listing 16.2.4.1:** Demographics

| | | | | | | | Specify | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Screening date | Sex | Date of birth (month/year) | Age | Ethnicity | other ethnicity | FAS | PP | Safety |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | PAT_FIRSTVISITDATE | PAT_GENDER | PAT_BIRTH_MONTH<br>PAT_BIRTH_YEAR | PAT_AGEYEAR | PAT_ETHNIC | PAT_ETHNIC_SP | [Derived data] | [Derived data] | [Derived data] |
| 04-CA-001 | Patient | 11/03/2011 | Male | 03/1959 | 54 | Other | XXXXXXXX | Yes | Yes | No |
| 04-CA-002 | Control | 09/04/2011 | Female | 09/1945 | 68 | Caucasian | | No | Yes | Yes |
| 04-CA-003 | Control | 10/07/2011 | Female | 02/1954 | 59 | Asian | | Yes | No | Yes |

Data Source Table: W\_PATIENT.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **50 of 167** 

### Listing 16.2.4.2: Carotid Ultrasound

| | | | | Righ | nt Side | L | eft Side |
|---|---|---|---|---|---|---|---|
| | | Has patient | | | Echolucency/Echogenicity | | Echolucency/ Echogenicity |
| Subject ID | Subject group* | history of TIA? | Carotid ultrasound date | Carotid stenosis | Grade# | Carotid stenosis | Grade# |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | [Derived data] | CU_DATE | CU_STEN_R | CU_ECHO_R | CU_STEN_L | CU_ECHO_L |
| 04-CA-001 | Patient | No | 11/03/2011 | 80% | 1 | 35% | 2 |
| 04-CA-002 | Control | No | 09/04/2011 | 35% | 3 | 58% | 4 |
| 04-CA-003 | Control | Yes | 10/07/2011 | 20% | 5 | 80% | 6 |

Data Source Table: W\_PATIENT, W\_CU, W\_MH.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>#</sup> Echolucency/Echogenicity grade: 1 = echolucent; 2 = predominantly echolucent; 3 = predominantly echogenic; 4 = echogenic




Version: 01 Page: **51 of 167** 

### **Listing 16.2.4.3:** Medical History and Associated Pathologies

| Subject ID | Subject group* | Medical condition | Preferred term | Date of diagnosis | Partial date | Ongoing? | Currently treated? | Resolution date | Partial date |
|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYP<br>E | MH_MEDCOND | MEDDRA_PT | MH_DIAGN_DATE | MH_PARTIAL_STAR<br>T_DATE | MH_ONGOING_YN | MH_TREATED_YN | MH_END_DATE | MH_PARTIAL_END_<br>DATE |
| 04-CA-001 | Patient | XXXXXX | XXXXXX | 15/08/1990 | Day | No | | 14/04/1994 | |
| 04-CA-002 | Control | XXXXXX | XXXXXX | 31/12/2007 | | No | | 15/06/2008 | Day&Month |
| 04-CA-003 | Control | XXXXXX | XXXXXX | 05/05/2005 | | Yes | Yes | | |

Data Source Table: W\_PATIENT, W\_MH.

Dictionary Name: MedDRA Version: 19.0

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **52 of 167** 

### **Listing 16.2.4.4/1: Prior and Concomitant Medications**

| | | Medication | ATC description | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | trade name | (third level) | Enrollment date | Start date | Partial date | Ongoing? | End date | Partial date |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | CM_NAME | ATC_LV3_DESC<br>R | PAT_FIRSTVISITDAT<br>E | CM_START_DATE | CM_PARTIAL_STAR<br>T_DATE | CM_ONGOING_YN | CM_END_DATE | CM_PARTIAL_END_<br>DATE |
| 04-CA-001 | Patient | XXXXXXX | XXXXXX | 11/03/2011 | 15/08/1990 | Day | No | 14/04/1994 | |
| 04-CA-002 | Control | XXXXXXX | XXXXXX | 09/04/2011 | 31/12/2007 | | No | 15/06/2008 | Day&Month |
| 04-CA-003 | Control | XXXXXXX | XXXXXX | 10/07/2011 | 05/05/2005 | | Yes | | |

Data Source Table: W\_PATIENT, W\_CM.

Dictionary Name: ATC Drug Dictionary Version: 2016

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **53 of 167** 

### **Listing 16.2.4.4/2: Prior and Concomitant Medications**

| | | Medication | ATC description | | | | Frequency of | Specify other | Route of | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | trade name | (third level) | Total daily dose | Unit | Specify other unit | administration | frequency | administration | Specify other route |
| PAT_PATNUMBE<br>R | PAT_INFCONS_T<br>YPE | CM_NAME | ATC_LV3_DESCR | CM_DOSE | CM_DOSEU | CM_DOSEU_SP | CM_FREQ | CM_FREQ_SP | CM_ROUTE | CM_ROUTE_SP |
| 04-CA-001 | Patient | XXXXXXX | XXXXXX | 3 | G | | BID | | Otherl | XXXXXX |
| 04-CA-002 | Control | XXXXXXX | XXXXXX | 3 | Other | XXXXXX | TID | | Intramuscolar | |
| 04-CA-003 | Control | XXXXXXX | XXXXXX | 12 | Mg | | Other | XXXXXX | Subcutaneous | |

Data Source Table: W\_PATIENT, W\_CM.

Dictionary Name: ATC Drug Dictionary Version: 2016

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **54 of 167** 

### Listing 16.2.5.1/1: Study Drug Administration and Extent of Subject Exposure

| - | Subject ID | Subject group* | Has the injection been performed? | Reason for not performing the injection | Injection date | Injection time | Batch of kit | Batch of<br><sup>99m</sup> Tc generator | _ |
|---|---|---|---|---|---|---|---|---|---|
| | PAT_PATNUMBER | PAT_INFCONS_TYPE | ANN_YN | ANN_YN_SP | ANN_DATE | ANN_TIME | ANN_KIT | ANN_GEN | |
| | 04-CA-001 | Patient | Yes | | 11/03/2011 | 10:50 | 09101-110631 | 09101-110631 | |
| | 04-CA-002 | Control | Yes | | 03/03/2011 | 10:00 | 09101-110981 | 09101-110981 | |
| | 04-CA-003 | Control | No | XXXXXXX | | | | | |

Data Source Table: W\_PATIENT, W\_ANN.

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **55 of 167** 

### Listing 16.2.5.1/2: Study Drug Administration and Extent of Subject Exposure

| | Subject ID | Subject group* | Has the injection been performed? | Radiochemical purity | Pre-injection total activity-dose in the syringe (MBq) | Post-injection residual activity-dose in the syringe (MBq) | Actual dose injected (MBq) | Volume of administered solution (mL) |
|---|---|---|---|---|---|---|---|---|
| - | PAT_PATNUMBER | PAT_INFCONS_TYPE | ANN_YN | ANN_TEST1 | ANN_TEST2_PRE | ANN_TEST2_POST | ANN_TEST2_EFF | ANN_TEST2_VOL |
| | 04-CA-001 | Patient | Yes | 98.7% | 123 | 123 | 123 | 123 |
| | 04-CA-002 | Control | Yes | 99.1% | 456 | 456 | 456 | 456 |
| | 04-CA-003 | Control | No | | | | | |

Data Source Table: W\_PATIENT, W\_ANN.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **56 of 167** 

### **Listing 16.2.6.1: Carotid and Aorta Imaging Assessment**

| | | Has patient | | Time from IP | Has the imaging | Reason for non | | | Have images been | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | history of TIA? | Imaging procedure | injection (min) | been completed? | completion | Date | Time | received and reviewed? | Result |
| PAT_PATNUMBE | PAT_INFCONS_TYP | [Derived data] | [Derived data] | [Derived data] | SP_YN | SP_YN_SP | SP_DATE | SP_TIME | SP_REV_YN | SP_RESULT |
| R | Е | [Delived data] | [Delived data] | [Derived data] | SPCT_YN | SPCT_YN_SP | SPCT_DATE | SPCT_TIME | SPCT_REV_YN | SPCT_RESULT |
| 04-CA-001 | Patient | No | SPECT | 60 | Yes | | 11/03/2011 | 10:50 | Yes | Positive |
| 04-CA-001 | Patient | No | SPECT/CT | 120 | Yes | | 11/03/2011 | 11:45 | Yes | Negative |
| 04-CA-002 | Control | No | SPECT | 60 | Yes | | 03/03/2011 | 10:00 | Yes | Negative |
| 04-CA-002 | Control | No | SPECT/CT | 120 | No | XXXXXX | | | | |

Data Source Table: W\_PATIENT, W\_MH, W\_SPECT\_SPECTCT.

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **57 of 167** 

## Listing 16.2.6.2: Carotid and Aorta Imaging Assessment – Uptake

| | | | | | Target to Background Ratio | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Has patient history of TIA? | Imaging procedure | Time from IP injection (min) | Left carotid | Right carotid | Thoracic aorta | Abdominal aorta | Aortic arch |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | [Derived data] | [Derived data] | [Derived data] | | | | | |
| 04-CA-001 | Patient | No | SPECT | 60 | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| 04-CA-001 | Patient | No | SPECT/CT | 120 | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| 04-CA-002 | Control | No | SPECT | 60 | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| 04-CA-002 | Control | No | SPECT/CT | 120 | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |

Data Source: Data provided by Sponsor.

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **58 of 167** 

### Listing 16.2.7.1/1: All Adverse Events

| | | | | Primary system | | | Study day of | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Event ID | Event description | organ class | Preferred term | Lowest level term | onset (days)§ | Ongoing? | Duration (days) | TEAE <sup>^</sup> | _ |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | MEDDRA_LLT | [Derived data] | AE_ONGOING_YN | [Derived data] | [Derived data] | |
| 04-CA-001 | Patient | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes | |
| 04-CA-002 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes | |
| 04-CA-003 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | Yes | YY | Yes | |

Note: NA = Not Available

^ TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>§</sup> Study day of onset is defined as days from Annexin injection



Version: 01 Page: **59 of 167** 

### Listing 16.2.7.1/2: All Adverse Events

| Subject ID | Subject group* | Event ID | Event description | AE caused<br>premature<br>withdrawal? | SAE | SAE seriousness | Maximal severity | Causal relationship with medication or procedure | Possible cause | Specify other possible cause | TEAE^ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TY<br>PE | ID_WEB | AE_NAME | AE_WITHD_YN | AE_SAE_YN | [Derived data] | AE_MAXSEV | AE_REL | AE_CAUSE | AE_CAUSE_SP | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | Yes | Yes | XXXXXX / XXXXX | Grade 2 (Moderate) | Possible | Other | XXXXXXXXX | Yes |
| 04-CA-002 | Control | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 1 (Mild) | Unlikely | Pre-existing/<br>underlying<br>disease | XXXXXXXXX | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 3 (Severe) | Unrelated | Other treatment | XXXXXXXXX | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1




Version: 01 Page: **60 of 167** 

### Listing 16.2.7.1/3: All Adverse Events

| Subject ID | Subject group* | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 04-CA-002 | Control | XXX | XXXXXXX | Dose modification in next treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1




Version: 01 Page: **61 of 167** 

### Listing 16.2.7.2/1: Serious Adverse Events

| | | | | Primary system | | | Study day of | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Event ID | Event description | organ class | Preferred term | Lowest level term | onset (days)§ | Ongoing? | Duration (days) | TEAE <sup>^</sup> | _ |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | MEDDRA_LLT | [Derived data] | AE_ONGOING_YN | [Derived data] | [Derived data] | |
| 04-CA-001 | Patient | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes | |
| 04-CA-002 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes | |
| 04-CA-003 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | Yes | YY | Yes | |

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

 $<sup>\</sup>S$  Study day of onset is defined as days from Annexin injection

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1





Version: 01 Page: **62 of 167** 

### Listing 16.2.7.2/2: Serious Adverse Events

| Subject ID | Subject group* | Event ID | Event description | AE caused premature withdrawal? | SAE | SAE seriousness | Maximal severity | Causal relationship with medication or procedure | Possible cause | Specify other possible cause | TEAE^ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TY<br>PE | ID_WEB | AE_NAME | AE_WITHD_YN | AE_SAE_YN | [Derived data] | AE_MAXSEV | AE_REL | AE_CAUSE | AE_CAUSE_SP | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | Yes | Yes | XXXXXX / XXXXX | Grade 2 (Moderate) | Possible | Other | XXXXXXXXX | Yes |
| 04-CA-002 | Control | XXX | XXXXXXXX | No | No | XXXXXX / XXXXX | Grade 1 (Mild) | Unlikely | Pre-existing/<br>underlying<br>disease | XXXXXXXXX | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 3 (Severe) | Unrelated | Other treatment | XXXXXXXXX | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1




Version: 01 Page: **63 of 167** 

### Listing 16.2.7.2/3: Serious Adverse Events

| Subject ID | Subject group* | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 04-CA-002 | Control | XXX | XXXXXXX | Dose modification in next treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1




Version: 01 Page: **64 of 167** 

### Listing 16.2.7.3/1: Adverse Events Leading to Withdrawal

| | | | | Primary system | | | Study day of | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Event ID | Event description | organ class | Preferred term | Lowest level term | onset (days)§ | Ongoing? | Duration (days) | TEAE^ |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | MEDDRA_LLT | [Derived data] | AE_ONGOING_YN | [Derived data] | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes |
| 04-CA-002 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes |
| 04-CA-003 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | Yes | YY | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Dictionary Name: MedDRA Version: XX.X

Note: NA = Not Available

^ TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>§</sup> Study day of onset is defined as days from Annexin injection



Version: 01 Page: **65 of 167** 

### Listing 16.2.7.3/2: Adverse Events Leading to Withdrawal

| Subject ID | Subject group* | Event ID | Event description | AE caused premature withdrawal? | SAE | SAE seriousness | Maximal severity | Causal relationship with medication or procedure | Possible cause | Specify other possible cause | TEAE^ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TY<br>PE | ID_WEB | AE_NAME | AE_WITHD_YN | AE_SAE_YN | [Derived data] | AE_MAXSEV | AE_REL | AE_CAUSE | AE_CAUSE_SP | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | Yes | Yes | XXXXXX / XXXXX | Grade 2 (Moderate) | Possible | Other | XXXXXXXXX | Yes |
| 04-CA-002 | Control | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 1 (Mild) | Unlikely | Pre-existing/<br>underlying<br>disease | XXXXXXXXX | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 3 (Severe) | Unrelated | Other treatment | XXXXXXXXX | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1




Version: 01 Page: **66 of 167** 

### Listing 16.2.7.3/3: Adverse Events Leading to Withdrawal

| Subject ID | Subject group* | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 04-CA-002 | Control | XXX | XXXXXXX | Dose modification in next treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1




Version: 01 Page: **67 of 167** 

### Listing 16.2.7.4/1: Adverse Events with Outcome Death

| | | | | Primary system | | | Study day of | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Event ID | Event description | organ class | Preferred term | Lowest level term | onset (days)§ | Ongoing? | Duration (days) | TEAE^ |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | MEDDRA_LLT | [Derived data] | AE_ONGOING_YN | [Derived data] | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes |
| 04-CA-002 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | No | YY | Yes |
| 04-CA-003 | Control | XXX | XXXXXX | XXXXXX | XXXXXXXX | XXXXXXX | YY | Yes | YY | Yes |

Note: NA = Not Available

^ TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>§</sup> Study day of onset is defined as days from Annexin injection



Version: 01 Page: **68 of 167** 

### Listing 16.2.7.4/2: Adverse Events with Outcome Death

| | | | Event | AE caused<br>premature | | | | Causal relationship with | | Specify other | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Event ID | description | withdrawal? | SAE | SAE seriousness | Maximal severity | medication or procedure | Possible cause | possible cause | TEAE <sup>^</sup> |
| PAT_PATNUMBER | PAT_INFCONS_TY<br>PE | ID_WEB | AE_NAME | AE_WITHD_YN | AE_SAE_YN | [Derived data] | AE_MAXSEV | AE_REL | AE_CAUSE | AE_CAUSE_SP | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | Yes | Yes | XXXXXX / XXXXX | Grade 2 (Moderate) | Possible | Other | XXXXXXXXX | Yes |
| 04-CA-002 | Control | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 1 (Mild) | Unlikely | Pre-existing/<br>underlying<br>disease | XXXXXXXXX | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 3 (Severe) | Unrelated | Other treatment | XXXXXXXXX | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1




Version: 01 Page: **69 of 167** 

### Listing 16.2.7.4/3: Adverse Events with Outcome Death

| Subject ID | Subject group* | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 04-CA-001 | Patient | XXX | XXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 04-CA-002 | Control | XXX | XXXXXXX | Dose modification in next treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 04-CA-003 | Control | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup> TEAE: Treatment Emergent Adverse Event as defined in paragraph 6.1.3.1





Version: 01 Page: **70 of 167** 

# Listing 16.2.8.1/1: Hematology

| Subject ID | Subject group* | Visit | Have hematology tests been done? | Sample collection<br>date | Sample collection time | Parameter | Result | Unit | Abnormality |
|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | VISIT_NAME | HE_YN | HE_DATE | HE_TIME | | HE_RBC | | HE_RBC_ABN |
| 04-CA-001 | Patient | Screening | Yes | 11/03/2011 | 10:52 | Red Blood Cells | 99.99 | 10 <sup>6</sup> /uL | Abnormal Non-Clinical Relevant |
| | | | | | | Hematocrit | 99.99 | % | Abnormal Non-Clinical Relevant |
| | | | | | | Etc. | 99.99 | | Abnormal Non-Clinical Relevant |
| 04-CA-001 | Patient | Visit 3 | Yes | 09/04/2011 | 15:00 | | 99.99 | | Abnormal Clinical Relevant |
| 04-CA-002 | Control | Screening | Yes | 10/07/2011 | 09:38 | | Not done | | |
| 04-CA-003 | Control | Visit 3 | No: XXXX | | | | | | |




Version: 01 Page: **71 of 167** 

Listing 16.2.8.2/1: Blood Chemistry

Repeat table 16.2.8.1 for Blood Chemistry parameters




Version: 01 Page: **72 of 167** 

Listing 16.2.8.3/1: Urinalysis

Repeat table 16.2.8.1 for Urinalysis parameters


#### **Statistical Analysis Plan ANNEXIN 04**


Version: 01 Page: **73 of 167** 

## Listing 16.2.8.4: Immunogenicity

| | | | Has venous | Reason for non | | | |
|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Visit | sample been done? | performance | Sample collection date | Sample collection time | _ |
| PAT_PATNUMBER | PAT_INFCONS_TYPE | VISIT_NAME | IM_YN | IM_YN_SP | IM_DATE | IM_TIME | |
| 04-CA-001 | Patient | Screening | Yes | | 11/03/2011 | 10:52 | |
| 04-CA-001 | Patient | Visit 3 | Yes | | 09/04/2011 | 15:00 | |
| 04-CA-002 | Control | Screening | Yes | | 10/07/2011 | 09:38 | |
| 04-CA-003 | Control | Visit 3 | No | XXXXXXXX | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IM. Other data source: database provided by Sponsor: XXXXXXXXX.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer



#### Statistical Analysis Plan ANNEXIN 04


Version: 01 Page: **74 of 167** 

# **Listing 16.2.9.1: Pregnancy Test**

| Subject ID | Subject group* | Sex | Age | Visit | Has the pregnancy test been performed? | Reason for non performance | Specify reason | Pregnancy test date | Pregnancy test time | Pregnancy test result |
|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | PAT_GENDER | PAT_AGEYEAR | VISIT_NAME | PT_YN | PT_NOTDONE | PT_NOTDONE_SP | PT_DATE | PT_TIME | PT_RESULT |
| 04-CA-001 | Patient | Male | 54 | Screening | Not applicable | | | | | |
| 04-CA-001 | Patient | Male | 54 | Visit 1 | Not applicable | | | | | |
| 04-CA-002 | Control | Female | 38 | Screening | Yes | | | 09/04/2011 | 12:00 | Negative |
| 04-CA-002 | Control | Female | 38 | Visit 1 | Yes | | | 12/04/2011 | 10:00 | Negative |
| 04-CA-003 | Control | Female | 59 | Screening | No | Menopause | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_PT.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **75 of 167** 

# **Listing 16.2.9.2:** Physical Examination

| | | | | | | | | | | Specify | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Visit | Evaluation period | Has physical examination been done? | Reason for non performance | Physical examination date | Physical examination time | Any clinically relevant finding? | First finding | Second finding | Third finding |
| PAT_PATNUMBE<br>R | PAT_INFCONS_<br>TYPE | VISIT_NAME | [Derived data] | PE_YN<br>PE_POST_YN | PE_YN_SP<br>PE_POST_YN_<br>SP | PE_DATE<br>PE_POST_DATE | PE_TIME<br>PE_POST_TIME | PE_RELFIND_YN<br>PE_POST_RELFI<br>ND_YN | PE_RELFIND1<br>PE_POST_RELFIN<br>D1 | PE_RELFIND2<br>PE_POST_RELFIN<br>D2 | PE_RELFIND3 PE_POST_RELFIN D3 |
| 04-CA-001 | Patient | Screening | | Yes | | 09/04/2011 | 12:00 | No | | | |
| 04-CA-001 | Patient | Visit 1 | Before injection | Yes | | 12/04/2011 | 10:00 | No | | | |
| 04-CA-001 | Patient | Visit 1 | After injection | Yes | | 12/04/2011 | 12:45 | Yes | XXXXX | XXXXXX | XXXXXX |
| 04-CA-002 | Control | Screening | | No | XXXXXXXX | | | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_PE\_VS, W\_PE\_VS\_POST.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **76 of 167** 

# Listing 16.2.9.3/1: Vital Signs

| | | | Evaluation | Have vital signs | Reason for | Vital signs | Vital signs | Systolic BP | Diastolic BP | Heart rate |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject group* | Visit | period | been evaluated? | non evaluation | evaluation date | evaluation time | (mmHg) | (mmHg) | (beats/min) |
| PAT PATNUMBER | PAT INFCONS TYPE | VISIT NAME | [Derived data] | VS_YN | VS_YS_SP | VS_DATE | VS_TIME | VS_SBP | VS_DBP | VS_HR |
| TAT_TATNOMBER | TAT_INI OONO_TTI L | VIOTI_IVAIVIL | [DCIIVOG Gata] | VS_POST_YN | VS_POST_YN_SP | VS_POST_DATE | VS_POST_TIME | VS_POST_SBP | VS_POST_DBP | VS_POST_HR |
| 04-CA-001 | Patient | Screening | | Yes | | 09/04/2011 | 12:00 | 165 | 99 | 77 |
| 04-CA-001 | Patient | Visit 1 | Before injection | Yes | | 12/04/2011 | 10:00 | 129 | 93 | 60 |
| 04-CA-001 | Patient | Visit 1 | After injection | Yes | | 12/04/2011 | 12:45 | 147 | 68 | 76 |
| 04-CA-002 | Control | Screening | | No | XXXXXXX | | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_PE\_VS, W\_PE\_VS\_POST.

Note: NA = Not Available

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer



Version: 01 Page: **77 of 167** 

# Listing 16.2.9.3/2: Vital Signs

| Subject ID | Subject group* | Visit | Has physical examination been done? | Reason for non performance | Physical examination date | Physical examination time | Height (cm) | Weight (Kg) | BMI (Kg/m^2) |
|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_INFCONS_TYPE | VISIT_NAME | PE_YN | PE_YN_SP | PE_DATE | PE_TIME | HEIGHT | WEIGHT | BMI |
| 04-CA-001 | Patient | Screening | Yes | | 09/04/2011 | 12:00 | 180 | 68.5 | 23.8 |
| 04-CA-002 | Control | Visit 1 | Yes | | 12/04/2011 | 10:00 | NA | 72.3 | 22.1 |
| 04-CA-003 | Control | Screening | Yes | | 06/05/2013 | 9:45 | 178 | 85.9 | 27.3 |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_PE\_VS.

Note: NA = Not Available

\* Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

# Statistical Analysis Plan ANNEXIN 04




Version: 01 Page: **78 of 167** 

# 11.2 Standard Tables





Version: 01 Page: **79 of 167** 

 Table 14.1.1:
 Subject Disposition

| POPULATION | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) | ALL SUBJECTS<br>(N=xx) |
|---|---|---|---|---|
| Screened subjects | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Screen failures | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Reason 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Reason m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Enrolled subjects | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Dosed subjects | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Completed study subjects | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Discontinued study subjects | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Reason 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Reason m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: All percentages are based upon the number of screened subjects.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer



#### Statistical Analysis Plan ANNEXIN 04


Version: 01 Page: **80 of 167** 

 Table 14.1.2:
 Analysis Populations

| ANALYSIS SET | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) | ALL SUBJECTS<br>(N=xx) |
|---|---|---|---|---|
| Full Analysis Set (FAS) | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Per Protocol population (PP) | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Safety population | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: All percentages are based upon the number of screened subjects.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **81 of 167** 

Table 14.1.3: Protocol Deviations

| PROTOCOL DEVIATION | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) | ALL SUBJECTS (N=xx) |
|---|---|---|---|---|
| Subjects with any minor protocol deviations | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Minor deviation 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Minor deviation m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Subjects with any major protocol deviations | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Major deviation 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Major deviation m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: All percentages are based upon the number of screened subjects.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **82 of 167** 

Table 14.1.4.1: Demographics – FAS Population

| PARAMETER | | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) | ALL SUBJECTS<br>(N=xx) |
|---|---|---|---|---|---|
| Age (years) | | n | 99 | 99 | 99 |
| | | Missing | 99 | 99 | 99 |
| | | Mean | 99.9 | 99.9 | 99.9 |
| | | S.D. | 99.9 | 99.9 | 99.9 |
| | | Median | 99.9 | 99.9 | 99.9 |
| | | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Sex | Male | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | Female | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Ethnicity | Asian | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | Black | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | Caucasian | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | Hispanic | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | Other | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: All percentages are based upon the number of enrolled subjects by group.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **83 of 167** 

## Table 14.1.5.1/1: Carotid Ultrasound – FAS Population

| RIGHT SIDE | | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|---|
| Carotid stenosis (%) | | n | 99 | 99 |
| | | Missing | 99 | 99 |
| | | Mean | 99.9 | 99.9 |
| | | S.D. | 99.9 | 99.9 |
| | | Median | 99.9 | 99.9 |
| | | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | | Min, Max | 99, 99 | 99, 99 |
| Echolucency/echogenicity grade | Echolucent | n (%) | 99 (99.9) | 99 (99.9) |
| | Predominantly echolucent | n (%) | 99 (99.9) | 99 (99.9) |
| | Predominantly echogenic | n (%) | 99 (99.9) | 99 (99.9) |
| | Echogenic | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: All percentages are based upon the number of enrolled subjects by group.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **84 of 167** 

## Table 14.1.5.1/2: Carotid Ultrasound – FAS Population

| LEFT SIDE | | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|---|
| Carotid stenosis (%) | | n | 99 | 99 |
| | | Missing | 99 | 99 |
| | | Mean | 99.9 | 99.9 |
| | | S.D. | 99.9 | 99.9 |
| | | Median | 99.9 | 99.9 |
| | | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | | Min, Max | 99, 99 | 99, 99 |
| Echolucency/echogenicity grade | Echolucent | n (%) | 99 (99.9) | 99 (99.9) |
| | Predominantly echolucent | n (%) | 99 (99.9) | 99 (99.9) |
| | Predominantly echogenic | n (%) | 99 (99.9) | 99 (99.9) |
| | Echogenic | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: All percentages are based upon the number of enrolled subjects by group.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **85 of 167** 

Table 14.1.6.1: Medical History and Associated Pathologies – Safety Population

| PRIMARY SYSTEM ORGAN CLASS PREFERRED TERM | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| Any medical and surgical history | n (%) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | n (%) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) |
| System organ class | n (%) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) |
| System organ class m | n (%) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Dictionary Name: MedDRA Version: XX.X

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **86 of 167** 

Table 14.1.7.1: Prior Medications or Non-Drug Therapies – Safety Population

| PHARMACOLOGICAL SUBGROUP<br>CHEMICAL SUBSTANCE | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| Any medication or therapy | n (%) | 99 (99.9) | 99 (99.9) |
| Pharmacological subgroup 1 | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance 1 | n (%) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance m | n (%) | 99 (99.9) | 99 (99.9) |
| Pharmacological subgroup | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance 1 | n (%) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance m | n (%) | 99 (99.9) | 99 (99.9) |
| Pharmacological subgroup m | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance 1 | n (%) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance m | n (%) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Dictionary Name: ATC Drug Dictionary Version: 2016

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one medication within a particular pharmacological subgroup and chemical substance will be counted only once for that pharmacological subgroup and chemical substance.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **87 of 167** 

Table 14.1.7.2: Prior and Concomitant Medications or Non-Drug Therapies – Safety Population

| PHARMACOLOGICAL SUBGROUP CHEMICAL SUBSTANCE | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| Any medication or therapy | n (%) | 99 (99.9) | 99 (99.9) |
| Pharmacological subgroup 1 | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance 1 | n (%) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance m | n (%) | 99 (99.9) | 99 (99.9) |
| Pharmacological subgroup | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance 1 | n (%) | 99 (99.9) | 99 (99.9) |
| ••• | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance m | n (%) | 99 (99.9) | 99 (99.9) |
| Pharmacological subgroup m | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance 1 | n (%) | 99 (99.9) | 99 (99.9) |
| ••• | n (%) | 99 (99.9) | 99 (99.9) |
| Chemical substance m | n (%) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Dictionary Name: ATC Drug Dictionary Version: 2016

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one medication within a particular pharmacological subgroup and chemical substance will be counted only once for that pharmacological subgroup and chemical substance.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer



Version: 01 Page: **88 of 167** 

## Table 14.1.8.1/1: Study Drug Administration – Safety Population

| QUALITY CONTROL ON<br>THE FINAL PRODUCT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| Radiochemical purity (%) | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: Acceptance criteria is radiochemical purity ≥ 90%.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **89 of 167** 

# **Table 14.1.8.1/2:** Study Drug Administration – Safety Population

| QUALITY CONTROL ON<br>THE FINAL PRODUCT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| Pre-injection total activity-dose in the syringe (MBq) | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| Post-injection residual activity-dose in the syringe (MBq) | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **90 of 167** 

# **Table 14.1.8.1/3:** Study Drug Administration – Safety Population

| QUALITY CONTROL ON<br>THE FINAL PRODUCT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| Actual dose injected (MBq) | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| Volume of administered solution (mL) | n | 99 | 99 |
| , , | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **91 of 167** 

Table 14.2.1.1: Carotid and Aorta Imaging Assessment – Prevalence of Positive Scans – FAS Population

| TIME POINT | | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|---|
| 60 mins after IP injection | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | 95% C.I. | 99.9 - 99.9 | 99.9 - 99.9 |
| | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| 120 mins after IP injection | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | 95% C.I. | 99.9 - 99.9 | 99.9 - 99.9 |
| | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| Overall# | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | 95% C.I. | 99.9 - 99.9 | 99.9 - 99.9 |
| | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Notes: All percentages are based upon the number of enrolled subjects by group.

Confidence intervals are estimated using the exact (Clopper-Pearson) formula for binomial proportions.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>#</sup> Subjects with either a positive scan at 60 or 120 minutes post injection will be considered overall positive





Version: 01 Page: **92 of 167** 

Table 14.2.1.2: Carotid and Aorta Imaging Assessment – Prevalence of Positive Scans – PP Population

| IMAGING PROCEDURE | | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|---|
| SPECT (60 mins after IP injection) | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | 95% C.I. | 99.9 - 99.9 | 99.9 - 99.9 |
| | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| SPECT/CT (120 mins after IP injection) | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | 95% C.I. | 99.9 - 99.9 | 99.9 - 99.9 |
| | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| Overall# | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | 95% C.I. | 99.9 - 99.9 | 99.9 - 99.9 |
| | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Notes: All percentages are based upon the number of enrolled subjects by group.

Confidence intervals are estimated using the exact (Clopper-Pearson) formula for binomial proportions.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>#</sup> Subjects with either a positive scan at 60 or 120 minutes post injection will be considered overall positive





Version: 01 Page: **93 of 167** 

Table 14.2.1.3: Patient Carotid and Aorta Imaging Assessment – Comparison between time points – FAS Population

| 60 MINS AFTER IP INJECTION | 120 MINS AFTER IP INJECTION | STATISTIC | PATIENT*<br>(N=xx) |
|---|---|---|---|
| Positive | Positive | n (%) | 99 (99.9) |
| Positive | Negative | n (%) | 99 (99.9) |
| Positive | Total | n (%) | 99 (99.9) |
| Negative | Positive | n (%) | 99 (99.9) |
| Negative | Negative | n (%) | 99 (99.9) |
| Negative | Total | n (%) | 99 (99.9) |
| Total | Positive | n (%) | 99 (99.9) |
| Total | Negative | n (%) | 99 (99.9) |
| Total | Total | n (%) | 99 (99.9) |
| | | p-value | 0.9999 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Notes: All percentages are based upon the number of subjects who performed both imaging procedures.

p-value is based on McNemar's test.

<sup>\*</sup> Patient = Subject with asymptomatic plaque





Version: 01 Page: **94 of 167** 

Table 14.2.1.4: Left Carotid Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population

| TIME POINT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| 60 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |
| 120 mins after IP injection | n | 99 | 99 |
| • | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

^p-value is based on T- test.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **95 of 167** 

Table 14.2.1.5: Right Carotid Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population

| TIME POINT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| 60 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |
| 120 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

^p-value is based on T- test.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **96 of 167** 

Table 14.2.1.6: Thoracic Aorta Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population

| TIME POINT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| 60 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |
| 120 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\* \*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer ^p-value is based on T- test.





Version: 01 Page: **97 of 167** 

Table 14.2.1.7: Abdominal Aorta Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population

| TIME POINT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| 60 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |
| 120 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

^p-value is based on T- test.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **98 of 167** 

Table 14.2.1.8: Aortic Arch Uptake Imaging Assessment – Target to Background Ratio (TBR) – FAS Population

| TIME POINT | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) |
|---|---|---|---|
| 60 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |
| 120 mins after IP injection | n | 99 | 99 |
| | Missing | 99 | 99 |
| | Mean | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 |
| | p-value^ | | 0.9999 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>^</sup>p-value is based on T-test.





Version: 01 Page: **99 of 167** 

Table 14.2.1.9: Left Carotid Uptake Imaging Assessment by ultrasound grade of plaque echolucency/echogenicity – Target to Background Ratio (TBR) – Patients - FAS Population

| TIME POINT | STATISTIC | ECHOLUCENT | PREDOMINANTLY<br>ECHOLUCENT | PREDOMINANTLY<br>ECHOGENIC | ECHOGENIC |
|---|---|---|---|---|---|
| 60 mins after IP injection | n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |
| 120 mins after IP injection | n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Patient = Subject with asymptomatic plaque

Only left carotid with stenosis >50% are taken into account.





Version: 01 Page: **100 of 167** 

Table 14.2.1.10: Right Carotid Uptake Imaging Assessment by ultrasound grade of plaque echolucency/echogenicity – Target to Background Ratio (TBR) – Patients - FAS Population

| TIME POINT | STATISTIC | ECHOLUCENT | PREDOMINANTLY<br>ECHOLUCENT | PREDOMINANTLY<br>ECHOGENIC | ECHOGENIC |
|---|---|---|---|---|---|
| 60 mins after IP injection | n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |
| 120 mins after IP injection | n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Patient = Subject with asymptomatic plaque

Only right carotid with stenosis >50% are taken into account.



#### Statistical Analysis Plan ANNEXIN 04


Version: 01 Page: **101 of 167** 

Table 14.3.1.1: Overall Summary of Adverse Events – Safety Population

| ADVERSE EVENT CATEGORY | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) | ALL SUBJECTS (N=xx) |
|---|---|---|---|---|
| Treatment emergent Aes | n (%) [n. events] | 99 (99.9) [99] | 99 (99.9) [99] | 99 (99.9) [99] |
| Treatment emergent adverse drug reactions | n (%) [n. events] | 99 (99.9) [99] | 99 (99.9) [99] | 99 (99.9) [99] |
| Treatment emergent SAEs | n (%) [n. events] | 99 (99.9) [99] | 99 (99.9) [99] | 99 (99.9) [99] |
| Treatment emergent serious adverse drug reactions | n (%) [n. events] | 99 (99.9) [99] | 99 (99.9) [99] | 99 (99.9) [99] |
| Treatment emergent AEs leading to withdrawal | n (%) [n. events] | 99 (99.9) [99] | 99 (99.9) [99] | 99 (99.9) [99] |
| Treatment emergent AEs leading to death | n (%) [n. events] | 99 (99.9) [99] | 99 (99.9) [99] | 99 (99.9) [99] |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: Format is number of subjects (percent of subjects) [number of events].

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **102 of 167** 

Table 14.3.1.2: Number (%) of Subjects Reporting Treatment Emergent Adverse Events by Primary System Organ Class and Preferred Term – Safety Population

| PRIMARY SYSTEM ORGAN CLASS<br>PREFERRED TERM | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) | ALL SUBJECTS<br>(N=xx) |
|---|---|---|---|---|
| Any adverse events | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary Name: MedDRA Version: 19.0

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **103 of 167** 

Table 14.3.1.3: Number (%) of Subjects Reporting Treatment Emergent Adverse Events by Severity – Safety Population

| PRIMARY SYSTEM ORGAN CLASS PREFERRED TERM | | Grade 1 Grad<br>(Mild) (Mode | | | | | Grade 4<br>(Threatening/<br>disabling) | | Grade 5<br>(Death) | | Mis | sing | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* |
| Any adverse events | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary Name: MedDRA Version: 19.0

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **104 of 167** 

Table 14.3.1.4: Number (%) of Subjects Reporting Treatment Emergent Adverse Drug Reactions by Severity – Safety Population

| PRIMARY SYSTEM ORGAN CLASS<br>PREFERRED TERM | Grade 1 Grad<br>(Mild) (Mode | | | | | Grade 4<br>(Threatening/<br>disabling) | | Grade 5<br>(Death) | | Missing | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* |
| Any adverse drug reactions | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary Name: MedDRA Version: 19.0

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **105 of 167** 

Table 14.3.1.5: Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Events by Primary System Organ

Class and Preferred Term – Safety Population

| PRIMARY SYSTEM ORGAN CLASS<br>PREFERRED TERM | STATISTIC | PATIENT*<br>(N=xx) | CONTROL*<br>(N=xx) | ALL SUBJECTS<br>(N=xx) |
|---|---|---|---|---|
| Any serious adverse events | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary Name: MedDRA Version: 19.0

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **106 of 167** 

Table 14.3.1.6: Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Events by Severity – Safety Population

| PRIMARY SYSTEM ORGAN CLASS<br>PREFERRED TERM | Grade 1 Grad<br>(Mild) (Mode | | | | | Grade 4<br>(Threatening/<br>disabling) | | Grade 5<br>(Death) | | Missing | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* |
| Any serious adverse events | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary Name: MedDRA Version: 19.0

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **107 of 167** 

Table 14.3.1.7: Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Drug Reactions by Severity – Safety Population

| PRIMARY SYSTEM ORGAN CLASS PREFERRED TERM | | | | de 2<br>erate) | | | Grade 4<br>(Threatening/<br>disabling) | | Grade 5<br>(Death) | | Missing | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* | Patient* | Control* |
| Any serious adverse drug reactions | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary Name: MedDRA Version: 19.0

Notes: All percentages are based upon the number of enrolled subjects by group.

Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer



#### **Statistical Analysis Plan ANNEXIN 04**


Version: 01 Page: **108 of 167** 

## Table 14.3.2.1: Listing of Adverse Events with Outcome Death – Safety Population

| Subject ID | Subject group* | Primary cause of death | Study drug injection date | Study drug injection time | Date of death | Time between study drug injection and death (days) | Relationship with study treatment |
|---|---|---|---|---|---|---|---|
| 04-CA-001 | Patient | Heart Attack | 10/05/2012 | 11:30 | 17/05/2012 | 7 | Probable |
| 04-CA-002 | Control | Aneurysm | 05/10/2012 | 12:38 | 08/10/2012 | 3 | Possible |
| 04-CA-003 | Control | Tuberculosis | 15/07/2012 | 09:45 | 16/10/2012 | 1 | Unlikely |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer


#### Statistical Analysis Plan ANNEXIN 04


Version: 01 Page: **109 of 167** 

#### Table 14.3.2.2: Listing of Serious Adverse Events – Safety Population

| Subject ID | Subject group* | Event description | Primary system<br>organ class | Preferred term | SAE date | Study day of onset (days)# | Duration<br>(days) | SAE criteria | Relationship with study treatment | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| 04-CA-001 | Patient | Vertigo | Ear and labyrinth disorders | Vertigo | 14/05/2012 | 1 | <1 | 2, 3 | Unlikely | Resolved |
| 04-CA-002 | Control | Fainting | Nervous system<br>disorders | Syncope | 10/09/2012 | 15 | <1 | 2 | Unlikely | Resolved with<br>sequelae |
| 04-CA-003 | Control | Internal<br>bleeding | Vascular disorders | Internal<br>haemorrhage | 16/11/2011 | 4 | 3 | 5 | Probable | Improved |
| | ••• | | ••• | ••• | | ••• | ••• | | ••• | |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary name: MedDRA Version 19.0

Note: SAE criteria: 1=Death, 2=Life-threatening, 3=Involved or prolonged hospitalization, 4=Congenital anomaly, 5=Persistent or significant disability or incapacity, 6=Significant from a medical standpoint.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>#</sup> Study day of onset is the day since Annexin administration which is defined as day 1.



#### **Statistical Analysis Plan ANNEXIN 04**


Version: 01 Page: **110 of 167** 

#### Table 14.3.4: Abnormal Laboratory Value Listing (Each Patient) – Safety Population

| Subject ID | Subject group* | Sex | Age | Dose of IP injected | Study day of onset (days)# | Laboratory<br>test type | Laboratory<br>test name | Laboratory<br>test value | Abnormal<br>non-clinically<br>relevant | Abnormal<br>clinical<br>relevant |
|---|---|---|---|---|---|---|---|---|---|---|
| 04-CA-001 | Patient | Male | 54 | 150 | 6 | Hematology | Red blood cells | 1000 | Yes | No |
| 04-CA-002 | Control | Female | 68 | 152 | 12 | Hematology | White blood cells | 1000 | No | Yes |
| 04-CA-003 | Control | Female | 59 | 150 | 26 | Blood chemistry | Gamma-GT | -54 | Yes | No |
| ••• | ••• | | | ••• | ••• | ••• | ••• | ••• | ••• | |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer

<sup>#</sup> Study day of onset is the day since Annexin administration which is defined as day 1.





Version: 01 Page: **111 of 167** 

## Table 14.3.5.1/1: Hematology – Red blood cells (10<sup>12</sup>/L) – Safety Population

| RED BLOOD CELLS (10^12/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **112 of 167** 

## Table 14.3.5.1/2: Hematology – Hematocrit (L/L) – Safety Population

| HEMATOCRIT (L/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **113 of 167** 

## Table 14.3.5.1/3: Hematology – Hemoglobin (g/L) – Safety Population

| HEMOGLOBIN (g/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **114 of 167** 

## Table 14.3.5.1/4: Hematology – White blood cells (10<sup>9</sup>/L) – Safety Population

| WHITE BLOOD CELLS (10^9/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **115 of 167** 

## Table 14.3.5.1/5: Hematology – Basophils (10<sup>9</sup>/L) – Safety Population

| BASOPHILS (10^9/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|--------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **116 of 167** 

## Table 14.3.5.1/6: Hematology – Eosinophils (10<sup>9</sup>/L) – Safety Population

| EOSINOPHILS (10^9/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|----------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **117 of 167** 

## Table 14.3.5.1/7: Hematology – Lymphocytes (10<sup>9</sup>/L) – Safety Population

| LYMPHOCYTES (10^9/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|----------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **118 of 167** 

## Table 14.3.5.1/8: Hematology – Monocytes (10<sup>9</sup>/L) – Safety Population

| MONOCYTES (10^9/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|--------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **119 of 167** 

## Table 14.3.5.1/9: Hematology – Neutrophils (10<sup>9</sup>/L) – Safety Population

| NEUTROPHILS (10^9/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|----------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **120 of 167** 

## Table 14.3.5.1/10: Hematology – Platelet Count (109/L) – Safety Population

| PLATELET COUNT (10^9/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **121 of 167** 

## Table 14.3.5.1/11: Hematology – PT (Second) – Safety Population

| PT (Second) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|-------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **122 of 167** 

# Table 14.3.5.1/12: Hematology – PTT (Second) – Safety Population

| PTT (Second) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|--------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **123 of 167** 

## Table 14.3.5.1/13: Hematology – INR – Safety Population

| INR | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|----------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **124 of 167** 

# Table 14.3.5.2/1: Blood Chemistry – ALP (U/L) – Safety Population

| ALP (U/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|-----------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **125 of 167** 

## Table 14.3.5.2/2: Blood Chemistry – ALT (U/L) – Safety Population

| ALT (U/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|-----------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **126 of 167** 

# Table 14.3.5.2/3: Blood Chemistry – AST (U/L) – Safety Population

| AST (U/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|-----------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **127 of 167** 

## Table 14.3.5.2/4: Blood Chemistry – Total Bilirubin (μmol/L) – Safety Population

| TOTAL BILIRUBIN (µmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **128 of 167** 

Table 14.3.5.2/5: Blood Chemistry – Direct Bilirubin (μmol/L) – Safety Population

| DIRECT BILIRUBIN (µmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **129 of 167** 

## Table 14.3.5.2/6: Blood Chemistry – Gamma-GT (U/L) – Safety Population

| GAMMA-GT (U/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|----------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **130 of 167** 

## Table 14.3.5.2/7: Blood Chemistry – Blood Urea Nitrogen (mmol/L) – Safety Population

| BLOOD UREA NITROGEN (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **131 of 167** 

## Table 14.3.5.2/8: Blood Chemistry – Albumin (g/L) – Safety Population

| ALBUMIN (g/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **132 of 167** 

Table 14.3.5.2/9: Blood Chemistry – Serum Creatinine (µmol/L) – Safety Population

| SERUM CREATININE (µmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **133 of 167** 

## Table 14.3.5.2/10: Blood Chemistry – Uric Acid (µmol/L) – Safety Population

| URIC ACID (µmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|--------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **134 of 167** 

## Table 14.3.5.2/11: Blood Chemistry – Sodium (mmol/L) – Safety Population

| SODIUM (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|-----------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **135 of 167** 

## Table 14.3.5.2/12: Blood Chemistry – Potassium (mmol/L) – Safety Population

| POTASSIUM (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|--------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **136 of 167** 

## Table 14.3.5.2/13: Blood Chemistry – Phosphorus (mmol/L) – Safety Population

| PHOSPHORUS (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **137 of 167** 

## Table 14.3.5.2/14: Blood Chemistry – Chloride (mmol/L) – Safety Population

| CHLORIDE (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|-------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **138 of 167** 

Table 14.3.5.2/15: Blood Chemistry – Corrected Calcium (mmol/L) – Safety Population

| CORRECTED CALCIUM (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **139 of 167** 

## Table 14.3.5.2/16: Blood Chemistry – Glucose (mmol/L) – Safety Population

| GLUCOSE (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **140 of 167** 

## Table 14.3.5.2/17: Blood Chemistry – Total Protein (g/L) – Safety Population

| TOTAL PROTEIN (g/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **141 of 167** 

## Table 14.3.5.2/18: Blood Chemistry – LDH (U/L) – Safety Population

| LDH (U/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|-----------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **142 of 167** 

## Table 14.3.5.2/19: Blood Chemistry – Total Cholesterol (mmol/L) – Safety Population

| TOTAL CHOLESTEROL (mmol/L) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **143 of 167** 

## Table 14.3.5.3/1: Urinalysis – Blood – Safety Population

| BLOOD | | | STATISTIC | SCREENING VISIT | VISIT 3 |
|---|---|---|---|---|---|
| Patient* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |
| Control* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **144 of 167** 

Table 14.3.5.3/2: Urinalysis – pH – Safety Population

| рН | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|----------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer




Version: 01 Page: **145 of 167** 

# Table 14.3.5.3/3: Urinalysis – Specific Gravity – Safety Population

| SPECIFIC GRAVITY | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|------------------|-----------|-----------------|------------|------------|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **146 of 167** 

# Table 14.3.5.3/4: Urinalysis – Protein – Safety Population

| PROTEIN | | | STATISTIC | SCREENING VISIT | VISIT 3 |
|---|---|---|---|---|---|
| Patient* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |
| Control* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **147 of 167** 

# Table 14.3.5.3/5: Urinalysis – Glucose – Safety Population

| GLUCOSE | | | STATISTIC | SCREENING VISIT | VISIT 3 |
|---|---|---|---|---|---|
| Patient* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |
| Control* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **148 of 167** 

# Table 14.3.5.3/6: Urinalysis – Ketones – Safety Population

| KETONES | | | STATISTIC | SCREENING VISIT | VISIT 3 |
|---|---|---|---|---|---|
| Patient* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |
| Control* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **149 of 167** 

## Table 14.3.5.3/7: Urinalysis – RBC (per high power field) – Safety Population

| RBC (PER HIGH<br>POWER FIELD) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **150 of 167** 

## Table 14.3.5.3/8: Urinalysis – WBC (per high power field) – Safety Population

| WBC (PER HIGH<br>POWER FIELD) | STATISTIC | SCREENING VISIT | VISIT 3 | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **151 of 167** 

Table 14.3.5.3/9: Urinalysis – Casts – Safety Population

| CASTS | | | STATISTIC | SCREENING VISIT | VISIT 3 |
|---|---|---|---|---|---|
| Patient* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |
| Control* | Test result | Negative | n (%) | 99 (99.9) | 99 (99.9) |
| | | Positive | n (%) | 99 (99.9) | 99 (99.9) |
| | | Not Done | n (%) | 99 (99.9) | 99 (99.9) |
| | | Missing | n (%) | 99 (99.9) | 99 (99.9) |
| | Change from baseline | Missing | n | - | 99 |
| | | Negative/Negative | n (%) | - | 99 (99.9) |
| | | Negative/Positive | n (%) | - | 99 (99.9) |
| | | Positive/Negative | n (%) | - | 99 (99.9) |
| | | Positive/Positive | n (%) | - | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **152 of 167** 

## Table 14.3.6.1/1: Vital Signs – Systolic Blood Pressure (mmHg) – Safety Population

| SYSTOLIC BLOOD<br>PRESSURE (mmHg) | STATISTIC | BASELINE | VISIT 1<br>(POST INJECTION) | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Baseline is the latest available assessment between screening and pre-injection visits.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **153 of 167** 

Table 14.3.6.1/2: Vital Signs – Diastolic Blood Pressure (mmHg) – Safety Population

| DIASTOLIC BLOOD<br>PRESSURE (mmHg) | STATISTIC | BASELINE | VISIT 1<br>(POST INJECTION) | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Baseline is the latest available assessment between screening and pre-injection visits.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer





Version: 01 Page: **154 of 167** 

## Table 14.3.6.1/3: Vital Signs – Heart Rate (beats/min) – Safety Population

| HEART RATE<br>(beats/min) | STATISTIC | BASELINE | VISIT 1<br>(POST INJECTION) | CHANGE |
|---|---|---|---|---|
| Patient* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |
| Control* | n | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Baseline is the latest available assessment between screening and pre-injection visits.

<sup>\*</sup> Patient = Subject with asymptomatic plaque; Control = Healthy volunteer






# 11.3 Standard Figures

The different lines on the figures should look different (e.g. dotted lines) rather than using different colours so that the lines can be distinguished when using a non-colour printer.



Version: 01 Page: **156 of 167** 

Figure 14.2.1.1: Left Carotid Target to Background Ratio (TBR) Imaging
Assessment - Patients - Carotid with Stenosis ≥ 50% - FAS
Population - 60 mins after IP injection





Version: 01 Page: **157 of 167** 







Version: 01 Page: **158 of 167** 







Version: 01 Page: **159 of 167** 







Version: 01 Page: **160 of 167** 







Version: 01 Page: **161 of 167** 







Version: 01 Page: **162 of 167** 







Version: 01 Page: **163 of 167** 







Version: 01 Page: **164 of 167** 







Version: 01 Page: **165 of 167** 





#### Statistical Analysis Plan ANNEXIN 04



Version: 01 Page: **166 of 167** 

#### 12 APPENDICES TO THE SAP TEMPLATE

## 12.1 Derived data

The following derived data will be calculated and included in the listings or in the tables:

### (1) Age

Subject age (years) will be derived as (informed conset date - birth date)/365.25 and truncated to the largest integer that is less than or equal to the calculated result. Since birth date is truncated (i.e. only month and year will be filled in the eCRF), it will be approximated using "01" as value for the day.

#### (2) **BMI**

BMI (kg/m²) will be automatically derived as [weight] (kg)/([height](cm)/100)² and rounded to the nearest decimal.

#### (3) Time from injection

Time from injection (min) will be derived as the difference between SPECT/CT scan time [SP\_TIME/SPCT\_TIME] and injection time [ANN\_TIME].

#### (4) Adverse event duration

If the start and end dates of the adverse event are identical then "<1" day will be presented with the duration in hh:mm recorded in the eCRF if it is available. If times are available, the duration will be calculated as (end date/time - start date/time) and presented in days hh:mm. If at least one time is missing and if the duration is greater than 24 hours then it will be calculated as (end date - start date)+1 and presented in days. If the recorded end date is CONT. (for continuing), the end date will be listed as "ongoing" and the duration will be approximated as "≥(last attended visit date - start date)+1" day(s). If the start date or the end date are partial the duration will be presented as a superior inequality "≥ xx" day(s) (i.e. "≥2" where start date = 31JAN2004 and end date = FEB2004 or start date = JAN2004 and end date = 01FEB2004).

#### (5) Study day of onset

If the start date of the adverse event is identical to the date of injection, then "1" day will be presented with the time to onset in hh:mm recorded in the eCRF if it is available. If the date of onset is greater than the date of injection then it will be calculated as (start date - injection date+1) and presented in days. If the date of onset precedes the date of injection the study day will be calculated as (start date - injection date). If the start date is partial, the time since injection will be presented as a superior

## Statistical Analysis Plan ANNEXIN 04




Version: 01 Page: **167 of 167** 

inequality (i.e. for an AE started in FEB2004 after the injection performed on 31JAN2004, the delay of onset will be "≥2" days).

## 12.2 SAS programs

This section provides the SAS programs related to the statistical tests specified in the statistical methods section 6. All computer output from SAS statistical programs used as a basis for extracted results should be retained for review by Responsible of statistical analysis.

| 4 | | | |
|---|--------|--------|-----------|
| 7 | 1 1212 | manır | NUITATION |
| | Dala | HIAHIL | ulation |

**Proc Format** 

**Proc Print** 

**Proc Sort** 

Proc SQL

**Proc Transpose** 

## 2 Descriptive statistics

Proc Corr

Proc Freq

**Proc Means** 

Proc Tabulate

#### 3 Test statistics

**Proc Ttest** 

## 4 Graphs

**Proc Boxplot** 

**Proc Sgplot**